## **CLINICAL TRIAL PROTOCOL**

A Multicenter, Open-Label, Flexible Dose Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients with Treatment-Resistant Childhood Absence Seizures

Protocol Number: INS011-17-113 Final Protocol Date: 23 Aug 2018

Version: 4.0

Investigational Product: Cannabidiol Oral Solution

IND Number: IND 123,120

ClinicalTrials.gov ID: NCT03355300

### CLINICAL TRIAL PROTOCOL

A Multicenter, Open-Label, Flexible Dose Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients with Treatment-Resistant Childhood Absence Seizures

Protocol Number: INS011-17-113

Protocol Date: 23 Aug 2018

Protocol Version: 4.0

Investigational Product: Cannabidiol Oral Solution

IND Number: 123,120

Sponsor: Insys Development Company, Inc.

1333 South Spectrum Blvd, Suite 100

Chandler, AZ 85286

Medical Monitor: PPD MD

Insys Development Company, Inc.

PPD Clinical Development

Phone: PPD

Fax: PPD

#### **Confidentiality Statement**

This study will be performed in compliance with Good Clinical Practices (GCP) and applicable regulatory requirements. The confidential information in this document is provided to you as an investigator, potential investigator or consultant for review by you, your staff and applicable Independent Ethics Committee (IEC) or Institutional Review Board (IRB). It is understood that the information will not be disclosed to others without written authorization from Insys Development Company, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

## PROTOCOL APPROVAL PAGE

A Multicenter, Open-label, Flexible Dose Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients with Treatment-Resistant Childhood Absence Seizures

## Protocol Approved by:

PPD PPD PPD Sr. Director, Clinical Operations Insys Development Company, Inc. Date: PPD PPD PPD Regulatory Affairs Date: 24 Auc 2018 Insys Development Company, Inc. PPD PPD MD PPD Clinical Development Insys Development Company, Inc.

### PROTOCOL SYNOPSIS

### Name of Sponsor/Company:

Insys Development Company, Inc.

## Name of Investigational Product:

Cannabidiol Oral Solution

## **Name of Active Ingredient:**

Cannabidiol

#### **Title of Study:**

A Multicenter, Open-label, Flexible Dose Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients with Treatment-Resistant Childhood Absence Seizures

Study center(s): Prospectively 8 sites will screen patients for enrollment

Phase of development: Phase 2 Long-Term Safety

## **Objective:**

The objective of this study is to assess the long-term safety and tolerability of Cannabidiol Oral Solution (CBD) in pediatric patients with treatment-resistant Childhood Absence Seizures.

#### Methodology:

This is a multicenter, open-label, flexible dose study designed to assess long-term safety and tolerability of CBD in doses ranging from 20 mg/kg/day to 40 mg/kg/day in patients with treatment-resistant childhood absence seizures. Patients must have completed INS011-17-103 to be eligible.

The Investigator will ensure that the patients legal representative [parent(s)/caregiver(s)] will receive a copy of the informed consent form for review and provide full informed consent prior to study participation. Patients may enroll in the Long-Term Safety study (INS011-17-113) after completing INS011-17-103 Visit 6 (End of Study) to avoid interruption of the investigational product. Patients will have up to 2 weeks to enroll in INS011-17-113. The first visit (Visit 1) for INS011-17-113 will be after the completion of Visit 6 of INS011-17-103.

Patients will continue to receive CBD treatment for approximately 48 weeks. Patients will remain on their previously assigned dose from Study INS011-17-103 or may be titrated up to a higher dose level if the Data Monitoring Committee (DMC) has approved the higher dose level in INS011-17-103. If any participant does not enroll within the 2 week window, that patient will not be eligible to enroll into the study.

The study will consist of a Safety Period (48±2 weeks), Taper Period (10±3 days), and a Follow-up Period (30±5 days). Treatment visits will be scheduled monthly for the first

3 months and then quarterly over the remaining 9 months. All patients will complete a Visit 7 (End of Study) or Early Withdrawal Visit regardless of when they stop treatment/complete the study. A Follow-Up telephone call (Visit 9) will occur 30 days after the end of either the End of Study (Visit 7) or Early Withdrawal.

In this study, all patients will be dosed as follows:

- Once the informed consent for INS011-17-113 is provided within the required time frame, initially the patient will receive the same dose as was administered during INS011-17-103. If tolerability issues occurred during INS011-17-103, the dose can be decreased if the dose was greater than 20 mg/kg/day. If the patient received 20 mg/kg/day and the physician wants to decrease the dose, the patient should be discontinued.
- Physicians will not increase a patient's assigned dose until the Data Monitoring Committee has deemed that the higher dose is safe in INS011-17-103. Doses of CBD may be adjusted at the investigator's discretion up to a maximum of 40 mg/kg/day.
- Treatment with established antiepileptic drugs (AEDs) and therapeutic treatments (e.g., vagus nerve stimulation [VNS]) may be initiated/continued/adjusted and changes will be permitted as necessary based on safety concerns or changes in seizure control. Any changes must be documented in the eCRF.

Patients will be dosed approximately every 12 hours with food to help ensure consistent plasma levels are achieved. Patients will be dosed for 48 weeks during which the investigator will assess safety and tolerability.

#### Study Assessments

At Visit 1 (Day 1) and each monthly and quarterly visit, the following assessments will be completed:

- Review of Antiepileptic Drugs (AEDs).
- Review of concomitant medications.
- Review of vital signs.
- Review clinical labs.
- Urinanalysis.

- Physical Examination (including height and weight).
- Brief Neurological Exam.
- Dispensing CBD.
- Drug Accountability.
- Review Adverse Events (AEs).
- 12-lead ECG.

At End of Study (Visit 7) or Early Withdrawal, the following assessments will be completed:

- Review of antiepileptic drugs (AEDs).
- Urinalysis.
- Urine pregnancy screen for postmenarchal females

- Review of concomitant medications.
- Review clinical labs
- 12-lead ECG.
- Review AEs.
- Review of vital signs
- Drug Accountability.

- Physical examination (including height and weight).
- Neurological examination
- Dispensing CBD.
- Columbia-Suicide Severity Rating Scale (C-SSRS).

At Taper Period (Visit 8), the following assessment will be completed:

- Collect CBD.
- Review AEs.

At Follow-Up (phone call only), the following assessments will be completed:

- Review of Antiepileptic Drugs (AEDs).
- Review of concomitant medications.
- Review AEs.

## Taper Period

At the end of the Long-Term Safety study, patients will be tapered off of CBD over a 0-10 days period. The following tapering scheme will be utilizied: 40 mg/kg/day will be reduced to 30 mg/kg/day for five days, then 20 mg/kg/day for five days, then stop; 30 mg/kg/day will be reduced to 20 mg/kg/day for five days, then stop; and doses  $\leq$  20 mg/kg/day can be discontinued without taper. This can be modified by the investigator based upon the patient's response.

Tapering will occur under the following circumstances:

- Patient completes Visit 7 (End of Study) of INS011-17-113
  - o Patient will begin tapering the day after Visit 7
- Patient withdraws early
  - o Patient will begin tapering the day after they decide to withraw from the trial

## Follow-Up Period

A Follow-up telephone call will occur 30 days after discontinuation of the study drug to assess AEs, AEDs, and record concomitant medications.

### **Number of patients (planned):**

Up to 30 patients who completed INS011-17-103 will be enrolled in the study.

### Diagnosis and main criteria for inclusion:

on 10/12/2022

#### Inclusion criteria

- 1. Completed activities up to and including Visit 6 (End of Study) of INS011-17-103.
- 2. Patient and/or parent(s)/caregiver(s) fully comprehend the informed consent form (ICF) and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
- 3. A female patient is eligible to participate in the study if she is:
  - a. Premenarchal, or
  - b. Of childbearing potential with a negative urine pregnancy test at the Screening Visit. If sexually active, she must agree to fulfill one of the following requirements:
  - i. Complete abstinence from intercourse for ≥ 4 weeks prior to administration of the first dose of the investigational product, throughout the Safety Period, and 4 weeks after completion or premature discontinuation from the investigational product, and agreement to use a double barrier method if she becomes sexually active.
  - ii. Use of acceptable methods of contraception throughout the study and 4 weeks after completion or premature discontinuation from investigational product. The acceptable method of contraception is double barrier method (i.e., condom plus spermicide or a condom plus intrauterine device [IUD], diaphragm, or stable hormonal contraceptive use for at least 3 months before screening and through 14 days after study completion).
- 4. A sexually active male patient or partner of enrolled patient must be willing to use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product. The acceptable methods of birth control are abstinence or double barrier birth control (i.e., condom plus spermicide or a condom plus one of the methods listed in criterion #3).
- 5. In the opinion of the investigator, the parent(s)/caregiver(s) is (are) willing and able to comply with the study procedures and visit schedules, including venipuncture, and the visit schedules.

#### Exclusion criteria

- 1. Patient or parent(s)/caregiver(s) have commitments during the study duration that would interfere with attending all study visits.
- 2. Experienced an anoxic episode related to study drug requiring resuscitation during the previous study.
- 3. Developed an adverse event thought to be related to CBD in the previous study and for whom the Investigator determines that continuing treatment with CBD would not be in the best interest of the patient.

- 4. Evidence of other clinically significant disease such as unstable hepatic, hematological, renal, cardiovascular, gastrointestinal, immunological, or pulmonary diseases or ongoing malignancies.
- 5. Compromised respiratory function or severe respiratory insufficiency.
- 6. Clinically significant abnormal laboratory values within the past 14 days, including:
  - a. Liver function tests (LFTs) such as albumin, direct bilirubin, total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≥3 times the upper limit of normal (ULN).
- 7. In the opinion of the investigator, the patient is unsuitable in any other way to participate in this study.

#### Investigational product, dosage and mode of administration:

Cannabidiol Oral Solution: an oral solution containing pharmaceutical grade synthetic cannabidiol manufactured and supplied by Insys Development Company, Inc.

Patients who completed INS011-17-103 will initiate this study on the dose with which they were receiving previously (20, 30, or 40 mg/kg/day orally). The total daily dose (mg/kg/day) will be administered in two equal doses (mg/kg) twice daily within 30 minutes after a meal. Doses of CBD may be adjusted at the investigator's discretion up to a maximum of 40 mg/kg/day once the higher dose level has been approved by the DMC in INS011-17-103.

Patients who withdraw early or complete this study will be tapered off in the following manner: 40 mg/kg/day will be reduced to 30 mg/kg/day for five days, then 20 mg/kg/day for five days, and then stop; 30 mg/kg/day will be reduced to 20 mg/kg/day for five days, then stop; and doses  $\leq$  20 mg/kg/day can be discontinued without taper. This can be modified by the investigator based upon the patient's response.

#### **Duration of treatment:**

The maximum duration of the study from Visit 1 (Day 1) to follow-up call will be approximately 54 weeks ( $\pm 3$  weeks).

### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

## Safety Endpoints

- Incidence, type, and severity of AEs and serious adverse events (SAEs) associated with Cannabidiol Oral Solution (i.e., treatment-emergent adverse events [TEAEs]).
- Changes from baseline in vital signs, ECG findings, and laboratory values (hematology, chemistry, and urinalysis).
- Changes from baseline in neurological exam.

Baseline is defined as Visit 6 of INS011-17-103.

#### **Statistical Methods:**

#### Safety Analysis

All safety assessments, including AEs, clinical laboratory evaluations, vital signs, 12-lead ECGs, physical examination (including height and weight), and neurological examinations will be listed for each visit. When appropriate, they will be summarized with descriptive statistics by age and dose cohort. The Medical Dictionary for Regulatory Activities (MedDRA; Version 20.0 or higher) will be used to classify all adverse events with respect to system organ class and preferred term. Adverse event summaries will include only TEAEs, which will be summarized for each treatment group.

- Clinical laboratory findings and vital signs will be summarized for all patients for observed values and change from baseline. Shifts from baseline to outside normal range criteria will also be presented for all patients.
- The neurological examination results will be listed and summarized descriptively. Shifts from baseline according to normal and abnormal criteria will also be presented for all patients.
- Results of physical examinations conducted throughout the study will be presented in listings and summarized descriptively. Shifts from baseline according to normal and abnormal criteria will also be presented for all patients.
- Concomitant medications and AEDs will be reported in the data listings.
- Statistical analyses will be performed using SAS® (Version 9.3 or higher, SAS Institute Inc.) or R (Version 3.3 or higher, Roswell Park Cancer Institute).

### **Missing Data**

There will be no imputation of the missing values. All assessments will be conducted based on all the observed data.

**Table 1:** Schedule of Events

| ASSESSMENTS | SAFETY PERIOD | | | | TAPER PERIOD | FOLLOW-UP<br>PERIOD <sup>i</sup> | |
|---|---|---|---|---|---|---|---|
| Visit Number | 1ª | 2, 3, 4<br>(monthly) | 5, 6<br>(quarterly) | 7<br>(End of Study) | Early<br>Withdrawal | 8 | 9<br>(Phone Call) |
| Study Time Points | Day 1 | Weeks 4, 8, 12 | Weeks 24, 36 | End of Active<br>Treatment (Week<br>48) | | 0-10 Days | 30 Days After EOS |
| Visit Window (Days) | ± 5 | ± 5 | ± 5 | ± 3 | | | ± 5 |
| Informed consent ** | | | | | | | |
| Review of inclusion/exclusion criteria ** | | | | 10 | | | |
| C-SSRS | | | | Х | X | | |
| Review of AEDs | X | X | Х | Х | X | | X |
| Review Concomitant<br>Medications | X | X | X | X | X | | X |
| Vital Signs <sup>b</sup> | X | X | X | X | X | | |
| Clinical Labs <sup>c</sup> | X | Х | Х | X | X | | |
| 12-lead ECG | X | X | X | X | X | | |
| Urinalysis | X | X | X | X | X | | |
| Urine pregnancy screen<br>for post-menarchal<br>females | X | | | X | X | | |
| Physical Examination <sup>d</sup> | X | X | X | X | X | | |
| Brief neurological<br>Examination <sup>e</sup> | X | X | X | X | X | | |
| Dosing with Cannabidiol<br>Oral Solution <sup>f</sup> | X | X | X | X | X <sup>f</sup> | Хg | |
| Drug Accountability | X | X | X | X | X | X | |
| AEs | X | X | X | X | X | X | X |

| ASSESSMENTS | SAFETY PERIOD | | | | TAPER PERIOD | FOLLOW-UP<br>PERIOD <sup>i</sup> | |
|---|---|---|---|---|---|---|---|
| Visit Number | 1ª | 2, 3, 4<br>(monthly) | 5, 6<br>(quarterly) | 7<br>(End of Study) | Early<br>Withdrawal | 8 | 9<br>(Phone Call) |
| Study Time Points | Day 1 | Weeks 4, 8, 12 | Weeks 24, 36 | End of Active<br>Treatment (Week<br>48) | | 0-10 Days | 30 Days After EOS |
| Visit Window (Days) | ± 5 | ± 5 | ± 5 | ± 3 | | | ± 5 |
| End of Study | | | | X | X <sup>h</sup> | | |

<sup>\*\*</sup> To be completed prior to enrollment into LTS, specifically within the 2 week period that is allotted post completion of Visit 6 (End of Study) of INS011-17-103.

<sup>i</sup> Follow-up Period visit (Visit 9) will be a phone call.

AE = adverse event; AED = anti-epileptic drug;

<sup>&</sup>lt;sup>a</sup> For patients who enroll within the first 2 weeks after completion of Visit 6 (End of Study) of INS011-17-103 protocol.

<sup>&</sup>lt;sup>b</sup> Vital signs will be taken after a 5-minute seated rest.

<sup>&</sup>lt;sup>c</sup> If the total bilirubin laboratory value is abnormal, direct bilirubin will be drawn.

<sup>&</sup>lt;sup>d</sup> The physical examination will include height, weight, and evaluation of general appearance, skin, eyes, ears, nose, throat, neck, lymph nodes, chest, heart, abdomen, and extremities.

e A brief neurological examination (mental status, cranial nerves, nystagmus, motor system, sensory system, reflexes, coordination, gait, and station) will be performed at all visits

<sup>&</sup>lt;sup>f</sup> At-home doses will be recorded in the daily medication diary.

g Following the Safety Period or if the patient withdraws early, the patient will enter a Taper Period. Patients will be tapered off of Cannabidiol Oral Solution as follows: 40 mg/kg/day will be reduced to 30mg/kg/day for five days, then 20 mg/kg/day for five days, then stop; 30 mg/kg/day for five days wil be reduced to 20 mg/kg/day for five days, then stop; 20 mg/kg/day can be discontinued without taper. This can be modified by the investigator based upon the patient's response.

h If the patient withdraws prematurely from the Safety Period, all Visit 7 (End of Study) procedures should be conducted. Site staff will follow up with the patient 4 weeks after completion of treatment via the telephone to collect information regarding AEs, AEDs, and concomitant medications.

# TABLE OF CONTENTS

| <b>PROTO</b> | COL APPROVAL PAGE | 2 |
|--------------|------------------------------------------------|----|
| PROTO | COL SYNOPSIS | 3 |
| TABLE | OF CONTENTS | 11 |
| List of 7 | Tables | 15 |
| List of F | Figures | 15 |
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 16 |
| 1. | INTRODUCTION | 19 |
| 1.1. | Cannabidiol | 19 |
| 1.1.1. | Mechanism of Action | 19 |
| 1.1.2. | Metabolism and Potential Drug Interactions | |
| 1.2. | Nonclinical Experience | 20 |
| 1.2.1. | Safety | 20 |
| 1.2.2. | Efficacy in Animal Models of Epilepsy | 20 |
| 1.3. | Clinical Experience. | |
| 1.3.1. | Overview of Safety | 23 |
| 1.3.2. | Pharmacokinetics | |
| 1.3.3. | Clinical Safety Data | 22 |
| 1.3.4. | Efficacy in Human Epilepsy | 25 |
| 1.4. | Childhood Absence Epilepsy | 25 |
| 1.5. | Dose Selection Rationale | 26 |
| 1.6. | Summary of Potential Risks and Benefits | 27 |
| 2. | STUDY OBJECTIVE | 29 |
| 3. | INVESTIGATIONAL PLAN | 30 |
| 3.1. | Overall Study Design | 30 |
| 3.1.1. | Safety Assessments | 31 |
| 3.1.2. | Taper Period | 31 |
| 3.1.3. | Follow-Up Period | 32 |
| 3.2. | Patient Selection | 32 |
| 3.2.1. | Inclusion Criteria | 32 |
| 3.2.2. | Exclusion Criteria | 32 |
| 3.3. | Removal of Patients from Therapy or Assessment | 35 |

| 3.4. | Dose Adjustment Criteria | 35 |
|----------|-----------------------------------------------------------|----|
| 3.5. | Stopping Rules | 36 |
| 4. | TREATMENTS | 37 |
| 4.1. | Treatments Administered | 37 |
| 4.2. | Identity of Investigational Product | 37 |
| 4.3. | Method of Assigning Patients to Treatment Groups | 37 |
| 4.4. | Selection and Timing of Dose for Each Patient | 37 |
| 4.5. | Blinding and Unblinding Treatment Assignment | 37 |
| 4.6. | Treatment Compliance | 37 |
| 4.7. | Permitted and Prohibited Therapies. | 38 |
| 4.7.1. | Permitted and Prohibited Therapies. Permitted Therapies. | 38 |
| 4.7.2. | Prohibited Therapies | 38 |
| 4.8. | Treatment After the End of Study | 38 |
| 5. | STUDY DRUG MATERIALS AND MANAGEMENT | 39 |
| 5.1. | Labeling and Packaging | 39 |
| 5.1.1. | Labeling | 39 |
| 5.1.2. | Packaging | 39 |
| 5.2. | Dispensing and Storage | 39 |
| 5.3. | Drug Supply and Accountability | 40 |
| 6. | STUDY ASSESSMENTS | 41 |
| 6.1. | Safety Assessments | 41 |
| 6.1.1. | Physical Examinations | |
| 6.1.2. | Neurological Examinations | 41 |
| 6.1.3. | Vital Signs | 41 |
| 6.1.4. | Electrocardiograms | 41 |
| 6.1.5. | Clinical Laboratory Assessments | 41 |
| 6.1.6. | Columbia Suicide Severity Rating Scale (C-SSRS) | 42 |
| 6.1.7. | Concomitant Medications | 42 |
| 6.1.8. | Adverse Events and Serious Adverse Events | 42 |
| 6.1.8.1. | Definition of Adverse Events | 42 |
| 6.1.8.2. | Classification of Adverse Events | 43 |
| 6.1.8.3. | Causality/Drug Relationship Assessment | 43 |
| 6.1.8.4. | Definition of Serious Adverse Events | 44 |

| 6.1.8.5. | Serious Adverse Events Actions Taken | 4 |
|---|---|---|
| 6.1.8.6. | Serious Adverse Events Outcome at the Time of Last Observation | 4 |
| 6.1.8.7. | Adverse Event Recording and Reporting | 4: |
| 6.1.8.8. | Adverse Event Follow-Up | 40 |
| 6.1.8.9. | Special Considerations | 40 |
| 7. | STUDY PROCEDURES | 4′ |
| 7.1. | Safety Period | 4′ |
| 7.1.1. | Visit 1 (Day 1) | 4′ |
| 7.1.2. | Monthly (Visits 2, 3, and 4) and Quarterly (Visits 5 and 6) Visits | 4′ |
| 7.2. | End of Study (Visit 7) or Early Withdrawal | 48 |
| 7.3. | Taper Period (Visit 8) | 48 |
| 7.4. | Follow-Up Period (Visit 9) | 48 |
| 8. | STATISTICS | 49 |
| 8.1. | STATISTICS Safety Endpoints | 49 |
| 8.2. | Sample Size Determination | |
| 8.3. | Analysis Populations | |
| 8.4. | Statistical Analyses | 49 |
| 8.4.1. | Study Patients and Demographics | 49 |
| 8.4.1.1. | Disposition and Withdrawals | 49 |
| 8.4.1.2. | Protocol Deviations | 49 |
| 8.4.1.3. | Demographics and Other Baseline Characteristics | 49 |
| 8.4.2. | Exposure and Compliance | 50 |
| 8.4.3. | Safety and Tolerability Analyses | 50 |
| 8.4.3.1. | Adverse Events | 50 |
| 8.4.3.2. | Clinical Laboratory Evaluations | 50 |
| 8.4.3.3. | Vital Signs | 50 |
| 8.4.3.4. | Electrocardiograms | 50 |
| 8.4.3.5. | Physical Examination Findings | 5 |
| 8.4.3.6. | Columbia Suicide Severity Rating Scale (C-SSRS) | 5 |
| 8.4.4. | Interim Analysis | 5 |
| 8.4.5. | Missing Data | 5 |
| 9. | STUDY CONDUCT | 52 |
| 9.1. | Sponsor and Investigator Responsibilities | 52 |

| 9.1.1. | Sponsor Responsibilities | 52 |
|---------|----------------------------------------------------|----|
| 9.1.2. | Investigator Responsibilities | 52 |
| 9.2. | Site Initiation | 53 |
| 9.3. | Screen Failures | 53 |
| 9.4. | Study Documents | 53 |
| 9.4.1. | Investigator's Regulatory Documents | 53 |
| 9.4.2. | Case Report Forms | 53 |
| 9.4.3. | Source Documents | 54 |
| 9.5. | Study Termination | 54 |
| 9.6. | Study Site Closure | 54 |
| 9.6.1. | Study Site Closure Record Retention | 54 |
| 9.6.2. | Laboratory Sample Retention | 55 |
| 10. | QUALITY CONTROL AND QUALITY ASSURANCE | 50 |
| 10.1. | Changes To The Protocol | 50 |
| 10.2. | Monitoring | |
| 10.3. | Data Review Meeting | 50 |
| 10.4. | Protocol Violations | 50 |
| 10.5. | Quality Assurance Audit | 5′ |
| 11. | REGULATORY AND ETHICAL CONSIDERATIONS | 58 |
| 11.1. | Regulatory Authority Approval | 58 |
| 11.2. | Ethical Conduct of the Study | 58 |
| 11.3. | Statement of Investigator/Delegation of Authority | 58 |
| 11.4. | Patient Informed Consent | 58 |
| 11.4.1. | Assent Guidance | 59 |
| 11.5. | Investigator Reporting Requirements | 59 |
| 12. | DATA HANDLING AND RECORD KEEPING | 60 |
| 12.1. | Data Management | 60 |
| 12.2. | Case Report Forms and Source Documents | 60 |
| 12.3. | Documentation and Retention of Essential Documents | 60 |
| 12.4. | Financial Disclosure | 60 |
| 13. | FACILITIES | 62 |
| 14. | USE OF INFORMATION AND PUBLICATION POLICY | 6. |
| 14.1. | Use of Information | 6 |

| Insys Deve | elopment Company, Inc. | Protocol Number INS011-17-113 |
|---|---|---|
| 14.2. | Publication Policy | 63 |
| 15. | REFERENCES (AVAILABLE UPON REQUEST | <sup>(</sup> )64 |
| 16. | INVESTIGATOR SIGNATURE PAGE | 67 |
| | List of Tables | |
| Table 1: | Schedule of Events | 9 |
| | List of Figures | |
| Figure 1: | Study Design Schematic | 33 |



## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

| Abbreviation or Specialist Term | Explanation |
|---|---|
| 5-HT <sub>1a</sub> | 5-hydroxytryptamine 1a |
| ACTH | adrenocorticotropic hormone |
| AE | adverse event |
| AEDs | anti-epileptic drugs |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| API | active pharmaceutical ingredient |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| AUC <sub>0-t</sub> | area under the concentration-time curve from 0 (predose) to |
| | the last quantifiable concentration |
| BMI | body mass index |
| BID | bis in die (twice a day) |
| BUN | blood urea nitrogen |
| CAE | childhood absence epilepsy1A1 |
| CB1 | cannabinoid receptor 1 |
| CB2 | cannabinoid receptor 2 |
| CBD | cannabidiol |
| CFR | Code of Federal Regulations |
| cGMP | current Good Manufacturing Practices |
| CLB | clobazam |
| C <sub>max</sub> | maximum plasma concentration |
| Ctrough | plasma trough concentrations |
| CNS | central nervous system |
| CRF | case report form |
| CRA | clinical research associate |
| CRO | contract research organization |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CV% | coefficient of variation |
| СҮР | cytochrome P450 |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| CYP1A1 | Cytochrome P450 1A1 |
| CYP2C19 | Cytochrome P450 2C19 |
| CYP2C9 | Cytochrome P450 2C9 |
| CYP3A4 | Cytochrome P450 3A4 |
| CYP3A5 | Cytochrome P450 3A5 |
| DEA | Drug Enforcement Administration |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EEG | electroencephalogram |
| EENT | eyes, ears, nose, and throat |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HIV | human immunodeficiency virus |
| IB | Investigator's Brochure |
| ICD | informed consent document |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Independent Ethics Committee |
| IFN | interferon |
| IL-2 | interleukin-2 |
| IP | Investigational product |
| IRB | Institutional Review Board |
| LDH | lactate dehydrogenase |
| MCT | medium chain triglycerides |
| MedDRA | Medical Dictionary for Regulatory Activities |
| ОН | hydroxy |
| PK | pharmacokinetic(s) |
| pKa | acid dissociation constant |
| PT | preferred term |
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|--------------------------------------|
| SOP | standard operating procedure |
| t½ | elimination half-life |
| TEAE | treatment-emergent adverse event |
| T <sub>max</sub> | time to maximum plasma concentration |
| $\Delta^9$ -THC | $\Delta^9$ -tetrahydrocannabinol |
| THC | tetrahydrocannabinol |
| US | United States |
| VNS | vagus nerve stimulation |



## 1. INTRODUCTION

Data presented in this section include overviews from the nonclinical and clinical published literature that reports on various other formulations of cannabidiol (CBD) (primarily plant-based). Analogous studies have not been completed for Cannabidiol Oral Solution, the synthetic pharmaceutical grade CBD to be investigated in this study.

Please see the Investigator's Brochure (IB)<sup>1</sup> for more information.

#### 1.1. Cannabidiol

The main active constituent of cannabis,  $\Delta^9$ -tetrahydrocannabinol ( $\Delta^9$ -THC) is the principal psychoactive constituent of marijuana. Cannabidiol is nonpsychoactive and the second most abundant cannabinoid. It has demonstrated a potential benefit to treating patients with treatment-resistant epilepsy.  $^{2,3,4,5}$ 

Insys Development Company, Inc. (hereafter referred to as the Sponsor) has successfully manufactured a pharmaceutical grade, synthetic CBD drug substance. It is manufactured in Insys' current Good Manufacturing Practices (cGMP) manufacturing facility. This facility is approved by the Drug Enforcement Administration (DEA) and has been inspected by the Food and Drug Administration (FDA). This active pharmaceutical ingredient is  $\geq 99.5\%$  pure<sup>6</sup> and can be consistently produced without concern for contaminant.

### 1.1.1. Mechanism of Action

The mode of action of CBD is not fully understood. The drug substance manifests a low affinity for endogenous cannabinoid receptors 1 (CB1) and 2 (CB2). Cannabidiol acts as an indirect antagonist of CB1 and inhibits several CB1 mediated  $\Delta^9$ -THC effects. It also stimulates the vanilloid receptor type  $1^8$  and modulates the  $\mu$ - and  $\delta$ -opioid receptors. It may also increase plasma  $\Delta^9$ -THC levels by inhibiting hepatic microsomal metabolism through competitively binding proteins in the cytochrome P450 (CYP) oxidative system. Finally, CBD may modulate neuronal hyperexcitability through one or more of the following mechanisms:

- Bidirectional regulation of calcium homeostasis via the mitochondrial sodium/calcium exchanger. 11
- Agonistic properties at 5-hydroxytryptamine 1a (5-HT<sub>1a</sub>) receptors. 12
- Enhancing endogenous adenosine levels in the central nervous system (CNS) by reducing adenosine re-uptake. 13,14

#### 1.1.2. Metabolism and Potential Drug Interactions

The major biotransformation pathway for CBD is similar to that of other cannabinoids and mediated by hydroxylation with cytochrome P450 (CYP) proteins. <sup>15</sup> Its interactions with human drug metabolizing enzymes (as a substrate, inhibitor, or inducer) were recently reviewed. <sup>16,17</sup>

Cannabidiol is metabolized primarily in the liver by CYP3A4 and to a lesser extent by CYP2C19. Specifically, CBD inhibits CYP3A4, CYP3A5, and CYP1A1 in vitro. 18,19,20 It also appears to inhibit CYP2C9<sup>21</sup> and the transport protein P-glycoprotein. 22,23

Further details may be found in the Investigator's Brochure (IB).<sup>1</sup>

23 Aug 2018

## 1.2. Nonclinical Experience

## **1.2.1.** Safety

In a nonclinical setting, single-dose toxicology studies of CBD reveal a relatively safe toxicology profile except at very high doses of the drug substance. Repeated dose toxicology studies highlight a potential impact of CBD on spermatogenesis, follicle-stimulating hormone levels, and a subset of immune responses.

Full detail of these results may be found in the IB.<sup>1</sup>

## 1.2.2. Efficacy in Animal Models of Epilepsy

Plant-derived CBD studies show antiepileptic,<sup>24</sup> antipsychotic, anti-dystonic, anti-emetic, and anti-inflammatory properties in animal models.<sup>25</sup> These models support exploring the use of CBD for the treatment of epilepsy.<sup>26</sup>

The anticonvulsant activity of oral CBD was investigated in an adult rat model of seizures (induced by maximal electroshock or audiogenic sources). Cannabidiol was effective against maximal electroshock-induced seizures (median effective dose  $[ED_{50}] = 18 \text{ mg/kg}$ ), but only minimally effective against audiogenic-induced seizures ( $ED_{50} \ge 75 \text{ mg/kg}$ ). The neurotoxicity median tolerated dose ( $TD_{50}$ ) was >100 mg/kg. Cannabidiol co-administered with different antiseizure drugs (e.g., phenytoin or carbamazepine) increased or reduced their anticonvulsant activity, indicating that synergism or antagonism with CBD was drug specific.

## 1.3. Clinical Experience

A Phase 1/2 study to assess the pharmacokinetics (PK) and safety of multiple doses (10 mg/kg/day, 20 mg/kg/day, and 40 mg/kg/day) of pharmaceutical grade, synthetic Cannabidiol Oral Solution in 61 pediatric patients with treatment-resistant seizure disorders aged 1 year to 17 years has been completed by the Sponsor (Protocol INS011-14-029). Patients were exposed for a period of approximately 11 days before qualifying to participate in the long-term extension study (INS011-14-030). Analyses demonstrated that:

- Cannabidiol levels on Day 10 appeared to increase proportionally with weight-based dose across the dosing cohorts, notwithstanding the two different formulations of the investigational product.
- Steady-state levels of cannabidiol appeared to be attained with approximately 2 to 6 days of repeated BID dosing with Cannabidiol Oral Solution, with geometric mean area under the concentration-time curve in plasma during a dosing interval (AUC<sub>(0-tau)</sub>) of 507.0 (Cohort 1 [10 mg/kg/day]), 836.0 (Cohort 2 [20 mg/kg/day]), and 2108 ng·h/mL (Cohort 3 [40 mg/kg/day]) for all age categories combined.
- Geometric mean maximum plasma concentrations (C<sub>max</sub>) of cannabidiol at steady-state were 91.0 (Cohort 1 [10 mg/kg/day]), 126.0 (Cohort 2 [20 mg/kg/day]), and 314.5 ng/mL (Cohort 3 [40 mg/kg/day]) for all age categories combined.
- Median time to maximum plasma concentration of cannabidiol at steady-state ranged from 2.0 to 3.0 hours for all age categories combined.

- Geometric means of cannabidiol apparent terminal half-life (t<sub>1/2</sub>) ranged from 19.5 to 29.6 hours following a single dose of Cannabidiol Oral Solution for all age categories combined.
- Accumulation in cannabidiol exposures was approximately 3- to 4-fold for all age categories combined. Dosing cohort total geometric means ranged from 2.6 to 3.1 for accumulation ratio for C<sub>max</sub> and from 3.6 to 4.4 for accumulation ratio for AUC<sub>(0-tau)</sub>.
- Most of the dosing cohort's total variability in cannabidiol exposures after repeated dosing (Day 10) was lower than Day 1. Single and repeated administrations of Cannabidiol Oral Solution resulted in highly variable systemic exposures of cannabidiol.
- There were no apparent formulation-related differences observed in terms of  $t_{1/2}$ , dose-normalized exposures, and variability.
- There were no clear trends for age-related differences in cannabidiol exposures, but exposure in infants tended to be lower than that in children and adolescents, approximately half at the highest dose (40 mg/kg/day).
- Approximately 50% of subjects enrolled were receiving clobazam. Clobazam and cannabidiol have a reciprocal drug-drug interaction leading to the increased mean exposures of both cannabidiol (approximately 2.5-fold), and clobazam as well as norclobazam (approximately 3-fold) at the highest dose (40 mg/kg/day).
- No apparent gender differences were observed for cannabidiol pharmacokinetics (PK).
- Pharmacokinetic results for 7-hydroxy cannabidiol and its statistical evaluations generally reflected those observed for parent cannabidiol.
- There were no quantifiable levels  $\Delta^9$ -THC and 11-hydroxy- $\Delta^9$ -THC measured following cannabidiol dosing.
- All doses of the investigational product were generally well-tolerated, although dose-titration was not employed. Dose-dependent adverse events (AEs) that occurred in multiple dosing cohorts and increased as the dose of the investigational product increased included diarrhea, flatulence, weight increase, somnolence, and psychomotor hyperactivity. Events of somnolence were potentially also related to concomitant use of clobazam with the investigational product, but this was not formally investigated in this study.
- There were no clinically relevant differences in the AE profile among subjects in the infant, child, and adolescent age categories.
- Serious adverse events were reported rarely and were consistent with underlying disease or procedures.
- Although this was not designed as an efficacy study, parent(s)/caregiver(s) and investigators both reported notable reductions in severity of mental illness (Clinical Global Impression of Severity) and improvement in global subject status (Clinical Global Impression of Improvement).

• The average change in weekly seizure rates (seizures of all types) was variable across subjects, dosing cohorts, and over time. Although the mean change in the weekly rate of tonic seizures at the end of the study compared with baseline generally decreased in a potentially dose-dependent manner, no pattern was observed for the other types of seizures reported. It was thought that tonic seizures were most representative of seizure control in this study.

In addition, a long-term safety study (Protocol INS011-14-030) for subjects enrolled in the PK study above was recently completed. Fifty-two of 61 subjects from INS011-14-029 enrolled; 45 subjects completed the study. There were seven early termination subjects (two for withdrawal of consent, two for AEs of aggressions and sleepiness/irritability, one for the SAE of worsening seizures, one for lack of efficacy, and one subject with a genetic mutation died from systemic sepsis and multi-organ failure considered nonrelated). Overall, 91% of the subjects were taking doses greater than 20 mg/kg/day, with 38% of subjects tolerating 40 mg/kg/day. The most common drug-related AEs reported were anemia (5 subjects), somnolence (4 subjects), and weight increased (4 subjects). However, the weight increases ranged from a little over 2 lbs to approximately 7 lbs.

During the study, trough PK values were drawn and interim PK data for CBD and 7-OH CBD from Visit 5 (Week 4) to Visit 8 (Week 24) were analyzed. Dose-normalized mean trough CBD concentrations ranged from 11.9 to 16 (ng/mL)/(mg/kg), showing relatively stable levels for up to 6 months dosing Cannabidiol Oral Solution at various dose levels. After one month of dosing, there did not appear to be much accumulation, even though early accumulation had likely happened when compared with INS011-14-029 results. High variability in trough CBD concentrations was observed, but the extent of variability between visits was similar as reported in the previous 029 study.

An open-label study of Cannabidiol Oral Solution (20 mg/kg/day and 40 mg/kg/day) in pediatric subjects with infantile spasms refractory to ACTH and vigabatrin recently was halted due to futility (Protocol INS011-15-054) because only one out of nine patients achieved a complete response.

A food effect study of Cannabidiol Oral Solution in normal healthy adults (Protocol INS011-15-043) recently completed and the results are presented in the IB. Analysis demonstrated significantly higher CBD levels when administered with food.

INS011-16-093 evaluated the effect of food on the bioavailability of multiple test formulations of Cannabidiol Oral Solution: MCT Oil formulation (100 mg/mL), Sesame Seed Oil formulation (100 mg/ml), and alcohol-containing formulation (80 mg/mL). The Sesame Oil formulation was studied both after subjects were fed a high fat diet and after a fast; the other formulations were tested after a high-fat diet. CBD  $C_{max}$  was approximately 12.3-fold higher after administration of food compared to fasting. Comparing the Sesame Oil fasting levels to the fed formulations there was a 12.7-fold higher CBD  $C_{max}$  (MCT formulation) and 11.2-fold higher  $C_{max}$  (alcohol-containing formulation).

Clinical data described in the following sections were collected following administration of various extracts of CBD as oral solutions or solid formulations.

## 1.3.1. Overview of Safety

Clinical studies in various human populations indicate that CBD has a favorable side-effect profile. Doses as high as 1500 mg are well tolerated.<sup>28</sup> No significant reactions or serious adverse events (SAEs) have been reported across a wide range of dosages in both acute and chronic settings. Bergamaschi et al.<sup>17</sup> recently reviewed the safety of CBD in humans and examined 221 subjects across 21 studies. As detailed in the IB<sup>1</sup>, no significant safety issues were reported.

Regarding doses of CBD that have been examined in other studies, daily doses of 200 to 300 mg CBD (or potentially more) may be safe. <sup>2,29</sup> Clinical evaluation and therapeutic ranges of CBD doses have been reported to be between 10 and 1500 mg/day, with the majority of reports evaluating doses in the 300 to 600 mg/day CBD range. Furthermore, between 300 and 1500 mg have been used in humans without toxicity or SAEs. <sup>30,31,32</sup>

#### 1.3.2. Pharmacokinetics

Study INS011-14-029 is a Phase 1/2 study assessing the PK and safety of multiple doses of CBD. In this recently completed PK trial using synthetic CBD (Cannabidiol Oral Solution, Insys Development Company, Inc.), each cohort consisted of 20 pediatric subjects from 1 to 17 years of age who received 10 mg/kg/day, 20 mg/kg/day, or 40 mg/kg/day over a period of 10 days. Subjects were dosed as in-subjects for Day 1 through Day 8. Subjects were then offered the opportunity to be discharged on Day 8 with readmission on Day 10 and a final study visit on Day 11. Cohort 1 received a formulation containing alcohol; Cohorts 2 and 3 received the final alcohol-free formulation containing medium chain triglycerides (MCT) oil. It was designed to have three age groups consisting of infants (1-2 yrs: 5 subjects), children (2 to <12 yrs: 9 subjects), and adolescents (12 to <17 yrs: 6 subjects) in each cohort.

Single oral administration of CBD at 5, 10, 20 mg/kg per dose resulted in mean peak levels of about 59, 111, and 232 ng/mL, respectively, and terminal half-life value of about 17 to 29 hours. The PK of CBD in different age groups was comparable at each dose level. Steady-state seemed to be achieved within 2 to 4 days after daily dose of 10, 20, 40 mg/kg/day CBD, with typical steady-state peak levels of about 120, 214, and 427 ng/mL, respectively, and a terminal half-life of 4 to 9 hours on Day 10.

Dose proportional increases in CBD exposures on Day 10 was clearly observed in mean  $C_{max,ss}$  and  $AUC_{tau}$  even if two different formulations were used in the study. Accumulation after repeated doses was about 2-fold. Plasma levels of 7-hydoxy (7-OH) CBD were generally similar to the parent drug.

Cannabidiol and clobazam (CLB) appear to have a drug-drug interaction based on the observed plasma levels of both drugs: Increase in mean exposures of clobazam on Day 10 by cannabidiol was shown in a dose-dependent matter (×1.2, × 1.5, × 2.6 of clobazam for 10, 20, 40 mg/kg/day CBD, respectively). Similarly, mean N-desmethyl CLB plasma levels following 20 or 40 mg/kg/day of CBD were increased by CBD.

However, there were appreciable changes in cannabidiol exposures on Day 10 only at the highest CBD dose (40 mg/kg/day), but not in the lower doses, with co-administration of clobazam.

The food effect study (Protocol INS011-15-043) demonstrated a 15 to 18-fold and 85-fold higher AUC and C<sub>max</sub>, respectively, in the fed state versus the fasting state after a single administration of 20 mg/kg Cannabidiol Oral Solution (300 mg/mL) in healthy adults. Inter-subject variability

was dramatically reduced with food: 55%CV from 125% for  $C_{max}$  and 35%CV from 78% for  $AUC_{0\text{-}inf}$ . Median time to maximum cannabidiol exposure ( $T_{max}$ ) occurred approximately 6 hours earlier under fed conditions compared to that after fasted conditions (6.00 h Fed vs. 12.00 h Fasted). The highest exposures with food in terms of AUC and  $C_{max}$  were 24040 h·ng/mL and 4190 ng/mL, respectively.

INS011-16-093 evaluated the effect of food on the bioavailability of multiple test formulations of Cannabidiol Oral Solution: MCT Oil formulation (100 mg/mL), Sesame Seed Oil formulation (100 mg/ml), and alcohol-containing formulation (80 mg/mL). The Sesame Oil formulation was studied both after subjects were fed a high fat diet and after a fast; the other formulations were tested after a high-fat diet. CBD  $C_{max}$  was approximately 12.3-fold higher after administration of food compared to fasting. Comparing the Sesame Oil fasting levels to the fed formulations there was a 12.7-fold higher CBD  $C_{max}$  (MCT formulation) and 11.2-fold higher  $C_{max}$  (alcohol-containing formulation).

As a comparison, mean peak and total exposures in all age groups (Protocol INS011-14-029) on Day 10 were within 16 to 36% to dose-adjusted exposures in fed adults (Protocol INS011-14-029).

#### 1.3.3. Clinical Safety Data

The following specific examples detail selected studies of the safety of CBD use in humans:

- Daily dosing of 10 mg/kg CBD was evaluated in a study of 15 subjects diagnosed with Huntington's disease.<sup>30</sup> Only 15 abnormal clinical laboratory values were associated with CBD treatment; these were largely limited to 4 subjects and exhibited no obvious pattern. No significant or clinical differences in CBD were observed in a cannabis-specific side-effect inventory.
- Chronic oral administration of 10 mg CBD daily for 21 days does not induce any changes in neurological (including electroencephalogram [EEG]), clinical (including electrocardiogram [ECG]), psychiatric, blood, or urine examinations in both healthy volunteers and epileptic subjects.<sup>2</sup>
- Oral administration of CBD in healthy volunteers (3 mg/kg daily for 30 days) and in epileptic subjects (200 to 300 mg daily for 135 days) was well tolerated. No signs of toxicity or serious side-effects were detected on neurological and physical examinations, blood and urine analysis, ECG, or EEG.<sup>2,29</sup>
- Administration of single and repeated doses of CBD for up to 20 days at a dose of 1200 mg/day does not impact pulse rate and blood pressure in human subjects with previous experience to cannabis smoking.<sup>34</sup>
- Three subjects with treatment-resistant schizophrenia have been dosed with 40 to 1280 mg/day of CBD for up to 4 weeks without reporting side-effects.<sup>35</sup>
- Two subjects diagnosed with bipolar affective disorder did not report adverse effects upon receiving 600 to 1200 mg/day of CBD for up to 24 days.<sup>36</sup>
- In addition, a long-term safety study (Protocol INS011-14-030) for subjects enrolled in the PK study above was recently completed. Fifty-two of 61 subjects from INS011-

14-029 enrolled; 45 subjects completed the study. There were seven early termination subjects (two for withdrawal of consent, two for AEs of aggressions and sleepiness/irritability, one for the SAE of worsening seizures, one for lack of efficacy, and one subject with a genetic mutation died from systemic sepsis and multi-organ failure considered nonrelated). Overall, 91% of the subjects were taking doses greater than 20 mg/kg/day, with 38% of subjects tolerating 40 mg/kg/day. The most common drug-related AEs reported were anemia (5 subjects), somnolence (4 subjects), and weight increased (4 subjects). However, the weight increases ranged from a little over 2 lbs to approximately 7 lbs.

## 1.3.4. Efficacy in Human Epilepsy

Several preliminary studies of CBD report reductions in seizure activity for a significant subset of subjects.

Plant-derived CBD was examined as an adjunctive therapy in 15 subjects with secondary generalized epilepsy with temporal focus who were refractory to conventional treatment.<sup>2,3</sup> The eight subjects randomized to the active arm received 200 to 300 mg/day of CBD or placebo for up to 4.5 months in addition to previously established antiepileptic drugs (AEDs).<sup>2,29</sup> Subjects tolerated CBD well, with no signs of toxicity or serious side-effects. Four of the eight subjects receiving CBD remained almost free of convulsive crises throughout the study and three others experienced partial improvement. The clinical condition of seven subjects receiving placebo remained unchanged and one subject improved.

Parents of children with treatment-resistant epilepsy have sought CBD-enriched cannabis for treatment.<sup>4</sup> In a survey, these parents reported dosages of CBD ranging from <0.5 to 28.6 mg/kg/day, as per results from medical cannabis testing facilities. Sixteen (84%) of the 19 parents eligible to respond to the survey reported a reduction in their child's seizure frequency while taking CBD-enriched cannabis. Of these, 2 (11%) reported complete seizure-freedom, 8 (42%) reported >80% reduction in seizure frequency, and 6 (32%) reported a 25% to 60% seizure reduction. Reported side-effects included fatigue and somnolence.

Realm Oil is an extract from a strain of cannabis known as Charlotte's Web and contains a CBD: $\Delta^9$ -THC ratio >20:1. Gedde and Maa<sup>5</sup> reported on a small group of pediatric subjects diagnosed with various types of epilepsy who took Realm Oil for  $\geq 3$  months. Baseline seizure frequency for these subjects ranged from 5 to 2800 events per week. Eight (8, 73%) of these subjects reported a 95% to 100% reduction in seizure occurrence, 1 (9%) reported 75% reduction, and 2 (18%) reported 20% to 45% reduction.

## 1.4. Childhood Absence Epilepsy

Although there are currently two drugs approved for childhood absence epilepsy (CAE), valproate and ethosuximide, neither are ideal. Valproate has potentially serious side effects, including weight gain, polycystic ovary disease, liver failure, and significant teratogenic effects. Ethosuximide does not control general tonic-clonic seizures that can co-exist with CAE. In a recent study comparing ethosuximide, valproic acid, and lamotrigine, freedom from failure rates where treatment failure was defined as persistence of absence seizures at Week 16 or 20, a generalized tonic-clonic seizure at any time, excessive drug-related systemic toxicity, dose-limiting toxicity after a single downward dose modification, or withdrawal initiated by the parent

or physician, was 53% (ethosuximide), 58% (valproic acid), and 29% (lamotrigine).<sup>37</sup> Therefore, there is still an unmet need for more effective anti-epileptic drugs with less side effects for these seizures. As CBD has been demonstrated to be effective in the treatment of cortical mediated epileptic encephalopathies,<sup>38</sup> Insys is proposing a multiple-site, open-label, dose-finding proof of concept study of Cannabidiol Oral Solution for the treatment of refractory childhood absence epilepsy.

#### 1.5. Dose Selection Rationale

Patients will initiate this long-term safety study on the final dose of Cannabidiol Oral Solution administered during the Phase 2 Study INS011-17-103.

Patients will not increase their assigned dose until the Data Monitoring Committee has approved the higher dose level in INS011-17-103. Doses of CBD may be adjusted at the investigator's discretion up to a maximum of 40 mg/kg/day.

## 1.6. Summary of Potential Risks and Benefits

As reviewed in Section 1.2 and Section 1.3, numerous nonclinical and clinical studies have examined other formulations of CBD. Several areas of potential concern have been identified with the use of CBD, especially in nonclinical studies. These include:

- Competitive binding of CYP proteins (thus, an impact on drug metabolism in the liver). Cannabidiol is metabolized predominantly by CYP3A4 and CYP 2C19.
   Cannabidiol may inhibit these 2 isozymes, as well as having small effects on CYP3A5, CYP1A1, and CYP2C9.
- Potential downregulation of immune responses involving the T, B, T-helper, and T cytotoxic subsets of leukocytes and/or those dependent on IL-2 or IFN-γ.

Based on recent studies of cannabinoid administration in humans, controlled CBD may be safe in humans and animals. However, further studies are needed to clarify these reported in vitro and in vivo side-effects.<sup>39</sup>

The inclusion/exclusion criteria, concomitant medication guidelines, and safety monitoring (AEs, clinical laboratory, vital signs, ECG, and physical examination assessments) planned for this study are intended to minimize these potential safety risks.

Criteria for removal of patients from the study will dictate discontinuation of patient participation should a safety issue arise (see Section 3.3).

Two facets of the current treatment landscape for pediatric patients with treatment-resistant absence seizures support the potential benefit for patients in this study. First, pediatric patients with treatment-resistant absence seizures continue to experience a significant unmet medical need despite ongoing treatment with currently available medications and procedures. Patients included in this study may potentially benefit from treatment with Cannabidiol Oral Solution. Devinsky et al.<sup>40</sup> recently noted that pediatric patients with treatment-resistant seizures are particularly good candidates for CBD intervention. Data reviewed in Section 1.2.2 and Section 1.3.4 demonstrate that CBD has shown preliminary efficacy in treating epilepsy in several early-stage nonclinical and clinical studies, respectively. This study is expected to serve as a critical step in the development of Cannabidiol Oral Solution as a treatment for refractory childhood absence epilepsy.

Second, synthetic pharmaceutical grade Cannabidiol Oral Solution is expected to have several distinct advantages over cannabis plant-derived extracts:

- Availability of the drug substance does not depend on cannabis plant production. As such, the development of Cannabidiol Oral Solution will not support growth and distribution of plants from which marijuana is derived.
- Manufacture of Cannabidiol Oral Solution does not involve an extraction process whereby the derived constituents could also include a significant amount of Δ<sup>9</sup>-THC. The manufacturing process can be controlled so that mass quantities can be produced that are uniform in quality, purity, and consistency and can be delivered in known and predetermined quantities.
- Variability in concentration and constituents should be reduced among batches, which may improve safety and tolerability.

• Reduced concern for contamination by  $\Delta^9$ -THC, herbicides, pesticides, etc.



#### 2. **STUDY OBJECTIVE**

The objective of this study is to assess the long-term safety and tolerability of Cannabidiol Oral Solution (CBD) in pediatric patients with treatment-resistant Childhood Absence Seizures.



## 3. INVESTIGATIONAL PLAN

## 3.1. Overall Study Design

This is a multicenter, open-label, flexible dose study designed to assess the long-term safety and tolerability of CBD in doses ranging from 20 mg/kg/day to 40 mg/kg/day in patients with treatment-resistant childhood absence seizures. Patients must have completed INS011-17-103 to be eligible.

The Investigator will ensure that the patients legal representative [parent(s)/caregiver(s)] will receive a copy of the informed consent form for review and provide full informed consent prior to study participation.

Patients should enroll in Long-Term Safety Study (INS011-17-113) after completing Study INS011-17-103 Visit 6 (End of Study) to avoid interruption of the investigational product. Patients will have up to 2 weeks to enroll in INS011-17-113. The first visit (Visit 1) for INS011-17-113 will be after the completion of Visit 6 of INS011-17-103.

Patients will continue to receive CBD treatment for approximately 48 weeks. Patients will remain on their assigned dose or may be titrated up to a higher dose level if the Data Monitoring Committee has approved the higher dose level in INS011-17-103. If any participant does not enroll within the 2 week window, the patient will not be eligible to enroll into the study.

The study will consist of a Safety Period (48±2 weeks), Taper Period (10±3 days), and a Follow-up Period (30±5 days). Treatment visits will be scheduled monthly for the first 3 months and then quarterly over the remaining 9 months. All patients will complete a Visit 7 (End of Study) or Early Withdrawal Visit regardless of when they stop treatment/complete the study. A Follow-Up telephone call (Visit 9) will occur 30 days after the end of either the End of Study (Visit 7) or Early Withdrawal.

In this study, all patients will be dosed as follows:

- Once the informed consent for INS011-17-113 is provided within the required time frame, initially the patient will receive the same dose as was administered during INS011-17-103. If tolerability issues occurred during INS011-17-103, the dose can be decreased if the dose was greater than 20 mg/kg/day. If the patient received 20 mg/kg/day and the physician wants to decrease the dose, the patient should be discontinued.
- Physicians will not increase a patient's assigned dose until the Data Monitoring Committee has deemed that the higher dose is safe in INS011-17-103. Doses of CBD may be adjusted at the investigator's discretion up to a maximum of 40 mg/kg/day.
- Treatment with established antiepileptic drugs (AEDs) and therapeutic treatments (e.g., vagus nerve stimulation [VNS]) may be initiated/continued/adjusted and changes will be permitted as necessary based on safety concerns or changes in seizure control. Any changes must be documented in the eCRF.

Patients will be dosed approximately every 12 hours with food to help ensure consistent plasma levels are achieved. Patients will be dosed for 48 weeks during which the investigator will assess safety and tolerability.

The study will be terminated upon one of the following:

- The investigational product is successfully approved for marketing in the US.
- Sponsor elects to terminate INS011-17-113.
- The patient has received 48 weeks of treatment.

## 3.1.1. Safety Assessments

At Visit 1 (Day 1) and each monthly and quarterly visit, the following assessments will be completed:

- Review vital signs, clinical labs, ECG, urinalysis, and physical examination (including height and weight). Refer to Section 6.1.
- Review adverse events (AEs). Refer to Section 6.1.8.
- 12-lead ECG.
- Brief neurological exam. Refer to Section 6.1.2.

At Visit 7 (End of Study) or Early Withdrawal Visits the following assessments will be completed:

- Columbia-Suicide Severity Rating Scale (C-SSRS) will be used for children and adolesents aged 7 to 17 years, if appropriate. Refer to Section 6.1.6.
- Review vital signs, clinical labs, ECG, urinalysis, and physical examination (including height and weight). Refer to Section 6.1.
- Review AEs. Refer to Section 6.1.8.
- Brief neurological exam. Refer to Section 6.1.2.

All AEs that arise during the Safety, Taper, and Follow-up Periods will be documented. Overall, patient safety will be reviewed as described in Section 10.3.

### 3.1.2. Taper Period

At the end of the Long-Term Safety study patients will be tapered off of CBD over a 0-10 days period. The following tapering scheme will be utilizied: 40 mg/kg/day will be reduced to 30 mg/kg/day for five days, then 20mg/kg/day for five days; 30mg/kg/day will be reduced to 20mg/kg/day for five days; and doses  $\leq 20$  mg/kg/day can be discontinued without taper. This can be modified by the investigator based upon the patient's response

Tapering will occur under the following circumstances:

- Patient completes Visit 7 (End of Study) of INS011-17-113.
  - o Patient will begin tapering the day after Visit 7.
- Patient withdraws early.
  - o Patient will begin tapering the day after the investigatory has been informed of the decision to withdraw from the trial.

## 3.1.3. Follow-Up Period

A follow-up telephone call (Visit 9) will occur 30 days after the Visit 7 (End of Study) or Early Withdrawal to assess AEs, AEDs, and record concomitant medications.



Figure 1: Study Design Schematic



## 3.2. Patient Selection

#### 3.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria:

- 1. Completed all activities through Visit 6 (End of Study) of INS011-17-103.
- 2. Patient and/or parent(s)/caregiver(s) fully comprehend the informed consent form (ICF) and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
- 3. A female patient is eligible to participate in the study if she is:
  - a. Premenarchal, or
  - b. Of childbearing potential with a negative urine pregnancy test at the Screening Visit. If sexually active, she must agree to fulfill one of the following requirements:
    - i. Complete abstinence from intercourse for ≥ 4 weeks prior to administration of the first dose of the investigational product, throughout the Safety Period, and 4 weeks after completion or premature discontinuation from the investigational product, and agreement to use a double barrier method if she becomes sexually active.
    - ii. Use of acceptable methods of contraception throughout the study and 4 weeks after completion or premature discontinuation from investigational product. The acceptable method of contraception is double barrier method (i.e., condom plus spermicide or a condom plus intrauterine device [IUD], diaphragm, or stable hormonal contraceptive use for at least 3 months before screening and through 14 days after study completion).
- 4. A sexually active male patient or partner of enrolled patient must be willing to use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product. The acceptable methods of birth control are abstinence or double barrier birth control (i.e., condom plus spermicide or a condom plus one of the methods listed in criterion #3).
- 5. In the opinion of the investigator, the parent(s)/caregiver(s) is (are) willing and able to comply with the study procedures and visit schedules, including venipuncture, and the visit schedules.

#### 3.2.2. Exclusion Criteria

Patients will be excluded for any of the following:

- 1. Patient or parent(s)/caregiver(s) have daily commitments during the study duration that would interfere with attending all study visits.
- 2. Experienced an anoxic episode related to study drug requiring resuscitation during their previous study.

- 3. Developed an adverse event thought to be related to CBD in the previous study and for whom the Investigator determines that continuing treatment with CBD would not be in the best interest of the patient.
- 4. Evidence of other clinically significant disease such as unstable hepatic, hematological, renal, cardiovascular, gastrointestinal, immunological, or pulmonary diseases or ongoing malignancies.
- 5. Compromised respiratory function or severe respiratory insufficiency.
- 6. Clinically significant abnormal laboratory values within the past 14 days, including:
  - a. Liver function tests (LFTs) such as albumin, direct bilirubin, total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT)  $\geq$  3 times the upper limit of normal (ULN).
- 7. In the opinion of the investigator, the patient is unsuitable in any other way to participate in this study.

## 3.3. Removal of Patients from Therapy or Assessment

Patients will be allowed to discontinue their participation in the study at any time for any reason (withdrawal of consent). Furthermore, participation in this clinical study may be discontinued by the investigator or by the sponsor for any of the following reasons:

- Intolerable side effects of the study product.
- Changes in medical status or medical condition of the patient such that the investigator believes that patient safety will be compromised or that it would be in the best interest of the patient to stop treatment.
- Patient safety or welfare is at risk.
- Non-compliance with study visits, defined as failure to perform any portion of scheduled assessments or procedures.
- Any unforeseen event that in the opinion of the treating physician and/or the Principal investigator, will prevent the research participant from continuing in this study.
- Sponsor decides to stop the study.

In the event of a patient's withdrawal, the investigator will promptly notify the sponsor. Every effort will be made to complete the end-of-study assessments.

Should any patient choose to withdraw early from the study, they will be advised of the safety precautions to be taken and will be followed until resolution of any AE or until the unresolved AEs are judged by the investigator to have stabilized.

# 3.4. Dose Adjustment Criteria

Doses of CBD may be adjusted at the investigator's discretion up to a maximum of 40 mg/kg/day only if the Data Monitoring Committee has approved the higher dose level in INS011-17-103. Doses greater than 40 mg/kg/day are not allowed. All dose changes must be clearly documented in the eCRF.
Antiepileptic drugs (AEDs) or therapies (e.g., VNS and ketogenic diet) may be initiated, discontinued or dose adjusted as needed. Any changes must be documented in the eCRF.

### 3.5. Stopping Rules

The investigator reserves the right to terminate the study in the interests of patient safety and welfare. The Sponsor reserves the right to terminate the study at any time for administrative reasons.

Patients will also be discontinued from the study if they meet the following criteria:

- ALT or AST > 3 x ULN with (or the appearance of) fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia >5%
- ALT or AST > 8 x ULN
- ALT or AST > 5 x ULN for more than 2 weeks
- ALT or AST > 3 x ULN and bilirubin > 2 x ULN or INR > 1.5

For patients meeting the above criteria, the investigator will arrange for the patient to return to the investigational site as soon as possible (within 24 hours of notice of abnormal results) for repeat assessment of ALT, AST, bilirubin, and alkaline phosphatase (ALP), detailed history, and physical examination. Patients will be followed until all abnormalities have normalized (in the investigator's opinion) or returned to the baseline state. If the patient is unable to return to the investigational site, repeat assessments may be performed at a local laboratory.

#### 4. TREATMENTS

#### 4.1. Treatments Administered

Patients or parent/caregiver will be reminded how to measure, take their dose, and record their dose in the dosing diary when the IP is dispensed for the first time.

Total daily doses ranging from 20 mg/kg/day to 40 mg/kg/day will be administered with food, within 30 minutes after a meal, in two equivalent daily doses approximately every 12 hours.

# 4.2. Identity of Investigational Product

The active pharmaceutical ingredient (API) in Cannabidiol Oral Solution is a pharmaceutical grade synthetic CBD manufactured according to cGMP. It is an off-white to pale yellow resin or crystal substance that is soluble in several organic solvents with an acid dissociation constant (pKa) of 9.64. The solution is a clear, colorless to pale yellow-brown colored solution (CBD concentration of 100 mg/mL) filled into a 30 mL amber glass vial. More detailed information may be found in the IB. <sup>1</sup>

# 4.3. Method of Assigning Patients to Treatment Groups

Patients will be allocated to a dose of the investigational product based on their dosing in the previous study INS011-17-103.

# 4.4. Selection and Timing of Dose for Each Patient

Once the informed consent for INS011-17-113 is provided, patients will initiate this long-term safety study on the final dose of CBD administered during the study INS011-17-103 Visit 6 (End of Study). Subsequently, the dose may be increased to a maximum of 40 mg/kg/day only if the higher dose level has been approved by the Data Monitoring Committee in INS011-17-103.

Patients will take each dose approximately every 12 hours with food in order to ensure consistent plasma levels are achieved. The date and time of all investigational product administrations will be documented in the case report form (CRF).

# 4.5. Blinding and Unblinding Treatment Assignment

Not applicable. This is an open-label study.

# **4.6.** Treatment Compliance

The prescribed dosage, timing, and mode of administration of IP may not be changed except as directed by the investigator.

The investigator, a member of the investigational staff, or a hospital pharmacist must maintain an adequate record of the receipt and distribution of all study medication using the Drug Accountability Form. These forms must be available for inspection at any time.

All supplies of IP should be accounted for at the termination of the study and a written explanation provided for discrepancies. All used and unused supplies, and packaging materials are to be inventoried and returned to the Sponsor or a designee by the investigator. The

investigator is not permitted to return or destroy unused clinical drug supplies or packaging materials unless authorized by the Sponsor or a designee.

If the study is terminated, discontinued, suspended, or completed, all used and unused supplies of the investigational product may be destroyed via the use of a third-party vendor or be returned to the Sponsor or a designee after the final drug accountability check has been performed. A certificate of destruction will be provided to the Sponsor.

All regulations issued by the DEA concerning the accountability of Schedule I medications will be followed (e.g., prevention of diversion).

# 4.7. Permitted and Prohibited Therapies

#### 4.7.1. Permitted Therapies

Any medications (other than those excluded by the protocol, see Section 4.7.2) that the investigator considers necessary for a patient's welfare and will not interfere with the investigational product may be administered at the investigator's discretion.

#### 4.7.2. Prohibited Therapies

During the Safety, Taper, and Follow-up Periods, patients are not to receive the following:

- Any cannabinoids besides the study drug (cannabidiol,  $\Delta^9$ -THC, hemp oil, Realm Oil or marijuana).
- Phenytoin, fluvoxamine, carbamazepine, or St. John's Wort.
- Medications that are strong inhibitors/inducers/sensitive substrates with a narrow therapeutic index for CYP3A4, CYP2C9, or CYP2C19, with the exception of Valproic Acid.
- Any other investigational drug or investigational device.

Although they are not prohibited, patients taking concomitant medications may need to be monitored with special care to identify any AEs arising due to the potential for altered drug metabolism.

# 4.8. Treatment After the End of Study

After the Safety Period, patients will have their taper schedule initiated over a 0-10 days period.

#### 5. STUDY DRUG MATERIALS AND MANAGEMENT

# 5.1. Labeling and Packaging

#### 5.1.1. Labeling

The labels for the investigational product will contain all information according to regulatory requirements.

#### 5.1.2. Packaging

The investigational product will be supplied in 30 mL containers of a 100 mg/mL strength (i.e., 3000 mg per container).

| Non-proprietary or common name of drug product | Cannabidiol Oral Solution, 100 mg/mL |
|---|---|
| Dosage form | Oral solution |
| Strength | 100 mg/mL |

Please refer to the Cannabidiol Oral Solution IB<sup>1</sup> for additional information on the drug formulation.

The investigational product will be clearly marked according to FDA and/or ICH requirements regarding use for clinical study investigation only and will be labeled with the investigational product name, study reference number, storage conditions, and expiry date. It is the responsibility of the investigator to ensure that accurate accountability records are maintained throughout the study. Study center staff will dispense the investigational product according to the handling instructions.

# 5.2. Dispensing and Storage

IP will be stored at controlled room temperature (20 to 25 degrees Celsius, 68 to 77 degrees Fahrenheit) at the study centers.

Cannabis and its constituents (including CBD) are **Schedule I** controlled substances and subject to all applicable local and federal laws and regulations regarding these products. This includes security provisions for storing the controlled substances and for dispensing in a manner to prevent diversion. Additionally, the Sponsor or investigator must provide a statement of the quantity to be manufactured and the sources of the chemicals to be used or the substance.

The DEA regulations detail specific security requirements for storage of the investigational product. Licensed practitioners must store controlled substances in a "securely locked, substantially constructed cabinet" and must notify the DEA of the theft or significant loss of any controlled substances within one business day of discovering such loss or theft. Furthermore, all practitioners are prohibited from hiring employees who have been convicted of a drug-related felony or who have had a DEA registration denied or revoked.

Investigators are responsible for ensuring that all applicable licensures are in place and storage conditions are appropriate.

Doses of IP will be administered from the Schedule I-licensed study center.

The study centers are required to provide complete information, including case report forms (CRFs) and final outcomes, on all instances of addiction, abuse, misuse, overdose, drug diversion/drug accountability, discrepancies in amount of the clinical supplies of the investigational product, noncompliance, protocol violations, lack of efficacy, individuals lost to follow-up, and any other reasons why patients dropped out of the study.

# 5.3. Drug Supply and Accountability

The investigator, a member of the investigational staff, or a hospital pharmacist must maintain an adequate record of the receipt and distribution of all study medication using the Drug Accountability Form. These forms must be available for inspection at any time.

All supplies of Cannabidiol Oral Solution should be accounted for at the termination of the study and a written explanation provided for discrepancies. All unused supplies and packaging materials are to be inventoried and returned to the Sponsor or a designee by the investigator. The investigator is not permitted to return or destroy unused clinical drug supplies or packaging materials unless authorized by the Sponsor or a designee.

If the study is terminated, discontinued, suspended, or completed, all unused supplies of the investigational product may be destroyed via the use of a third-party vendor or be returned to the Sponsor or a designee after the final drug accountability check has been performed. A certificate of destruction will be provided to the Sponsor.

All regulations issued by the DEA concerning the accountability of Schedule I medications will be followed (e.g., prevention of diversion).

#### 6. STUDY ASSESSMENTS

# **6.1.** Safety Assessments

For all patients physical examination, brief neurological examination, vital signs (seated blood pressure, pulse rate, temperature, and respiration rate), clinical laboratory testing (hematology, chemistry, and urinalysis), 12-lead ECG, concomitant medication, C-SSRS, and AE assessments (including TEAEs and SAEs).

#### 6.1.1. Physical Examinations

A physical examination (evaluation of general appearance, skin, eyes, ears, nose, throat, neck, lymph nodes, chest, heart, abdomen, and extremities) will be conducted for every patient during the Visit 1 (Day 1), all monthly and quarterly visits, and Visit 7 (End of Study) or Early Withdrawal.

#### 6.1.2. Neurological Examinations

A brief neurological examination (mental status, cranial nerves, nystagmus, motor system, sensory system, reflexes, coordination, gait, and station) will be conducted for Visit 1 (Day 1), all monthly and quarterly visits, and Visit 7 (End of Study) or Early Withdrawal.

#### 6.1.3. Vital Signs

Vital signs (seated blood pressure, pulse rate, temperature and respiration rate) will be measured during Visit 1 (Day 1), all monthly & quarterly visits, and Visit 7 (End of Study) or Early Withdrawal. Additional vital sign measurements may be performed as deemed medically necessary by research personnel.

### 6.1.4. Electrocardiograms

A resting 12-lead ECG will be conducted for every patient at Visit 1 (Day 1), all monthly & quarterly visits, and Visit 7 (End of Study) or Early Withdrawal.

#### 6.1.5. Clinical Laboratory Assessments

Blood samples for hematology and chemistry assessments and urine sample for urinalysis will be collected during Visit 1 (Day 1), all monthly & quarterly visits, and Visit 7 (End of Study) or Early Withdrawal.

- Hematology: hemoglobin, hematocrit, total and differential leukocyte count, red blood cell (RBC), and platelet count.
- Chemistry: albumin, blood urea nitrogen (BUN), creatinine, total bilirubin, alkaline phosphatase (ALP), aspartate transaminase (AST), alanine transaminase (ALT), sodium (Na<sup>+</sup>), potassium (K<sup>+</sup>), chloride (Cl<sup>-</sup>), lactate dehydrogenase (LDH), uric acid, glucose, and calcium.
- Urinalysis: pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrite, leukocyte esterase, and urobilinogen. If protein, occult blood, nitrite, or leukocyte esterase values are out of range a microscopic examination will be performed.

A urine dipstick pregnancy test will be performed on all female post-menarchal patients during at Visit 1 and Visit 7 (End of Study) or Early Withdrawal.

#### 6.1.6. Columbia Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a prospective assessment tool routinely used in studies of drugs with any potential for CNS effects. It captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. For patients aged 7 to 17 years and if the developmental level is appropriate, the questionnaire will be completed at the end of the Safety Period (Visit 7) or Early Withdrawal. For patients who are less than 7 years or for whom the C-SSRS is inappropriate due to the patient's developmental functioning, a clinical assessment will be made following FDA guidelines.

(https://www.fda.gov/downloads/drugs/guidances/ucm225130.pdf).

Patients who have significant findings for suicidal ideation as assessed by the C-SSRS must be referred to the investigator for follow-up evaluation.

#### **6.1.7.** Concomitant Medications

Will be assessed at all visits.

#### 6.1.8. Adverse Events and Serious Adverse Events

#### **6.1.8.1.** Definition of Adverse Events

An AE is defined as any untoward medical occurrence in a patient administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product.

Patients will be monitored throughout the study for AEs. Monitoring for treatment-emergent AEs will begin as soon as the patient is dosed. All AEs must be followed until they are resolved or stabilized, or until all attempts to determine resolution of the event are exhausted. The investigator should use their discretion in ordering additional tests as necessary to monitor the progress of such events.

An AE may be:

23 Aug 2018

- A new illness, not documented in the patient's s medical history;
- Worsening of a concomitant illness;
- An effect of the study medication; it could be an abnormal laboratory value, as well as a significant shift from baseline within normal range which the qualified investigator or medical qualified designate considers to be clinically important;
- A combination of two or more of these factors.

Surgical procedures themselves are not AEs. They are therapeutic measures for conditions that required surgery. The condition for which the surgery is required is an AE, if it occurs or is detected during the study period. Planned surgical measures permitted by the clinical study protocol and the conditions(s) leading to these measures are not AEs, if the condition(s) was

(were) known before the start of study treatment. In the latter case, the condition should be reported as medical history.

Absence seizures will not be considered AEs. However, new seizure types and injury resulting from a seizure will be captured as AEs.

Patients will be monitored throughout the study for AEs. All AEs must be followed until they are resolved or stabilized, or until all attempts to determine resolution of the event are exhausted. The investigator should use his/her discretion in ordering additional tests as necessary to monitor the progress of such events.

Adverse events reported prior to dose administration will be recorded as part of the patient's medical history.

Previous clinical trial experience has shown that somnolence, diarrhea, and transaminase elevations may be associated with CBD treatment. Therefore, Insys Development Company has identified these as Adverse Events of Special Interest.

#### **6.1.8.2.** Classification of Adverse Events

Adverse events are to be recorded on the AE page of the patient's case report form (CRF). Severity will be graded according to the following definitions:

- <u>Mild</u>: The patient experiences awareness of symptoms but these are easily tolerated or managed without specific treatment.
- <u>Moderate</u>: The patient experiences discomfort enough to cause interference with usual activity, and/or the condition requires specific treatment.
- <u>Severe</u>: The patient is incapacitated with inability to work or do usual activity, and/or the event requires significant treatment measures.

Action taken will be categorized as none, study drug discontinued, dose modified, required concomitant medication, required procedure, or other.

Event outcome at resolution or time of last follow-up will recorded as event resolved, resolved with sequelae, ongoing, or death.

#### 6.1.8.3. Causality/Drug Relationship Assessment

The relationship of the event to the study drug should be determined by the investigator according to the following criteria:

- <u>Definitely related</u>: The event follows a reasonable temporal sequence from the time of drug administration that cannot be explained, follows a known or expected response pattern to the study drug, that is confirmed by improvement on stopping and reappearance of the event on repeated exposure and that could not be reasonably explained by other factors such as the patient's clinical condition, intercurrent illness, or concomitant drugs.
- Not related: The event is most likely produced by other factors such as the patient's clinical condition, intercurrent illness, or concomitant drugs, and does not follow a

known response pattern to the study drug, or the temporal relationship of the event to study drug administration makes a causal relationship unlikely.

- <u>Possibly related</u>: The event follows a reasonable temporal sequence from the time of drug administration, and/or follows a known response pattern to the study drug, but could have been produced by other factors such as the patient's clinical condition, intercurrent illness, or concomitant drugs.
- <u>Unlikely related</u>: The event follows little or no temporal sequence from the time of drug administration that makes a causal relationship improbable and/or other factors such as the patient's clinical condition, intercurrent illness, or concomitant drugs is a more likely alternative.
- <u>Probably related</u>: The event follows a reasonable temporal sequence from the time of drug administration, and/or follows a known response pattern to the study drug, and cannot be reasonably explained by other factors such as the patient's clinical condition, intercurrent illness, or concomitant drugs.

#### **6.1.8.4.** Definition of Serious Adverse Events

A serious AE (SAE) is any AE that fulfills any of the following criteria, as per 21 CFR 312.32:

- Results in death;
- Is life-threatening;
- Requires in-patient hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant disability or incapacity;
- Is a congenital anomaly or birth defect;
- Is medically significant or requires intervention to prevent one of the outcomes listed above.

Serious AEs will be captured from the time of consent through the end of the study.

#### 6.1.8.5. Serious Adverse Events Actions Taken

Actions taken may consist of:

- None: No action taken
- Treatment: Standard of care measures instituted
- Drug withdrawn: Study medication was permanently discontinued because of the AE
- Unknown: Not known, not observed, not recorded, or refused

#### 6.1.8.6. Serious Adverse Events Outcome at the Time of Last Observation

The outcome at the time of last observation will be classified as:

- Recovered/resolved
- Recovered/resolved with sequelae

- Not recovered/not resolved
- Death
- Unknown

#### 6.1.8.7. Adverse Event Recording and Reporting

Adverse events will be recorded throughout the study in the source documents and in the CRFs. The investigator will rate AEs for seriousness, intensity, causality, action taken, and outcome as described in the previous section.

Expedited reporting is required for serious unexpected adverse drug reactions. Fatal or life-threatening unexpected drug reactions must be reported by the Sponsor to regulatory agencies no more than 7 days after the Sponsor's first knowledge of the reaction; followed by as complete a report as possible within 8 additional days. Unexpected drug reactions must be reported no later than 15 days after the Sponsor's first knowledge of the reaction. In order to comply with these requirements, the investigator or delegate must inform the Sponsor immediately upon occurrence of any SAE. The site will complete the SAE Report Form as thoroughly as possible and e-mail it to Insys within 24 hours of the investigators first knowledge of the event.

Sponsor contact information is listed below:

### **Insys Development Company, Inc.**

Email: clinicalpv@insysrx.com

These SAE reports must contain the following information:

- A. Study name/number
- B. Study drug
- C. Investigator details (name, phone, fax, e-mail)
- D. Patient number
- E. Patient initials
- F. Patient demographics
- G. Clinical event
  - 1) Description
  - 2) Date of onset
  - 3) Treatment (drug, dose, dosage form)
  - 4) Adverse event relationship to study drug
  - 5) Action taken regarding study drug in direct relationship to the AE
- H. If the AE was fatal or life-threatening
- I. Cause of death (whether or not the death was related to study drug)

# J. Autopsy findings (if available)

The Sponsor or its representative will be responsible for notification to regulatory agencies.

### 6.1.8.8. Adverse Event Follow-Up

All non-serious AEs that are not related or unlikely to be related to study treatment will be followed until the end of study participation. All SAEs or AEs that are considered as possibly, probably, or definitely related to treatment will be followed until resolution or stabilization.

#### **6.1.8.9.** Special Considerations

Cannabidiol inhibits drug metabolism mediated by a subset of CYP proteins (see Section Section 1.1.2). Thus, the investigator and study center staff should monitor patients who are taking concomitant medications that are metabolized by CYP2C19, CYP2C9, CYP2D6, CYP3A4, CYP1A2, or by P-glycoprotein with special care.

#### 7. STUDY PROCEDURES

Prior to performing any study related procedures or assessments, the Investigator will ensure that the patients and/or their parent(s)/caregiver(s) (if applicable) provide written informed consent and that the perdiatric patient provides assent (as appropriate). Patients and their parent(s)/caregiver(s) (if applicable) will receive a copy of the informed consent form (ICF) and asent form for review and must provide fully informed consent prior to study participation.

The consent process must be conducted and the ICF signed before any study procedures. See Section 11.4 for guidelines regarding patient consent and assent.

The assessments and procedures that will be conducted during this study are summarized in Table 1.

### 7.1. Safety Period

# 7.1.1. Visit 1 (Day 1)

The following procedures and assessments will be performed:

- Review/Assess past/current AEDs and concomitant medications.
- Record vital signs, collect blood samples for clinical labs, and collect urine sample for urinalysis.
- Urine dipstick pregnancy test (all female patients of childbearing potential).
- Perform physical and <u>brief</u> neurological examinations.
- 12-lead ECG.
- Collect/review/dispense CBD (dose may be modified up to 40 mg/kg/day at investigator's discretion).
- Perform drug accountability.
- Review AEs.

# 7.1.2. Monthly (Visits 2, 3, and 4) and Quarterly (Visits 5 and 6) Visits

The following procedures and assessments will be performed:

- Review/Assess past/current AEDs and concomitant medications.
- Record vital signs, collect blood samples for clinical labs, complete 12-lead ECG, and collect urine sample for urinalysis.
- Perform physical and brief neurological examinations.
- Collect/review/dispense CBD (dose may be modified up to 40 mg/kg/day at investigator's discretion).
- Perform drug accountability.
- Review AEs.

# 7.2. End of Study (Visit 7) or Early Withdrawal

The following procedures and assessments will be performed:

- Review/assess past/current AEDs and concomitant medications.
- Record vital signs, collect blood samples for clinical labs, complete 12-lead ECG, and collect urine sample for urinalysis.
- Perform physical and <u>brief</u> neurological examinations.
- Collect/review CBD (dose may be modified up to 40 mg/kg/day at investigator's discretion).
- Perform drug accountability.
- Review AEs.
- Complete C-SSRS.
- Urine dipstick pregnancy test (all female patients of childbearing potential).
- Dispense CBD for Taper Period.
- End of Study assessments (If the patient withdraws prematurely from the Safety Period, all Visit 7 (End of Study) procedures should be conducted. Site staff will follow-up with the patient 4 weeks after completion of treatment via the telephone to collect information regarding AEs, AEDs, and concomitant medications.

# 7.3. Taper Period (Visit 8)

The following procedures and assessments will be performed:

- Collect CBD.
- Review AEs.

# 7.4. Follow-Up Period (Visit 9)

The following assessments will be performed by phone call 30 days after Visit 7 (End of Study) the last study dose:

- Review/assess past/current AEDs and concomitant medications.
- Review AEs.

#### 8. **STATISTICS**

#### 8.1. **Safety Endpoints**

Changes in safety endpoints will be reported as mean/median change from baseline at relevant time points and as a listing of events that fall outside normal limits. Baseline is defined as Visit 6 of INS011-17-103.

- Incidence, type, and severity of AEs and serious adverse events (SAEs) associated with Cannabidiol Oral Solution (i.e., treatment-emergent adverse events [TEAEs]).
- Changes from baseline in vital signs, physical exam (including height and weight), ECG findings, and laboratory values (hematology, chemistry, and urinalysis).
- Changes from baseline in neurological exam.

#### 8.2. **Sample Size Determination**

The sample size is based on successful completion of INS011-17-103, with a maximum of 30 patients.

#### **Analysis Populations** 8.3.

Statistical analysis will be conducted on all enrolled patients.

#### 8.4. **Statistical Analyses**

This section presents a summary of the planned statistical analyses. A Statistical Analysis Plan (SAP) that describes the details of the analyses to be conducted will be finalized prior to database lock.

Summary statistics will be provided for the variables described as follows. For continuous variables, these statistics will typically include the number of patients, mean, standard deviation, median, minimum, and maximum. For categorical variables, these statistics will typically include the number and percentage of patients in each category.

#### 8.4.1. **Study Patients and Demographics**

# **8.4.1.1.** Disposition and Withdrawals

The numbers of patients entering, completing, and withdrawing, along with reasons for withdrawal, will be tabulated overall and by modal dose group. For each patient, the modal dose is the dose with the longest exposure during the study.

#### **8.4.1.2.** Protocol Deviations

23 Aug 2018

Protocol deviations will be identified and classified as minor or major and listed.

# 8.4.1.3. Demographics and Other Baseline Characteristics

Demographic and baseline characteristics (including age, gender, race, weight, height, and BMI) will be summarized by for the overall population by descriptive statistics. No formal statistical

49

analyses will be performed. Medical history, clinical laboratory test results, and ECG assessments will be listed and summarized by descriptive statistics.

Prior and concomitant medications will be summarized by the number and percentage of patients taking each medication. They will also be classified by using the World Health Organization Drug Dictionary Anatomical Therapeutic Chemical classes and preferred terms.

# **8.4.2.** Exposure and Compliance

The exposure to study medication will be summarized by descriptive statistics. Any compliance deviations will be listed.

# 8.4.3. Safety and Tolerability Analyses

No formal inferential analyses will be conducted for safety variables. Data listings will be provided for protocol-specified safety data.

### 8.4.3.1. Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA, version 20.0 or higher) will be used to classify all AEs. Adverse event summaries will include only TEAEs, which will be summarized for each modal dose group. For each patient, the modal dose is the dose with the longest exposure during the study.

The number and percentage of patients with AEs will be displayed for each treatment group by system organ class and preferred term. Summaries of AEs by severity and relationship to the IP will also be provided. Serious AEs (SAEs) and AEs resulting in discontinuation will be summarized separately in a similar manner. Patient listings of AEs and SAEs will be produced.

# 8.4.3.2. Clinical Laboratory Evaluations

For the continuous laboratory parameters, descriptive statistics will be presented for values collected at all study visits as indicated in Table 1.

# **8.4.3.3.** Vital Signs

For blood pressure, pulse rate, temperature, and respiration rate, descriptive statistics will be presented for values collected at all study visits as indicated in Table 1.

# 8.4.3.4. Electrocardiograms

For the continuous ECG parameters, descriptive statistics will be presented for values collected at each visit, and for the changes from Baseline to End of Study/Early Withdrawal.

Additionally, the number and percentage of patients will be presented as shift tables for the overall interpretation from Screening (normal or abnormal, not clinically significant [NCS]) to End of Study/Early Withdrawal (normal; abnormal, NCS; or abnormal, clinically significant [CS]).

# **8.4.3.5.** Physical Examination Findings

Physical examination body systems will be presented as the number and percentage of patients that have normal or abnormal results at each visit. The examination will include evaluation of height, weight, general appearance, skin, eyes, ears, nose, throat, neck, lymph nodes, chest, heart, abdomen, and extremities.

# 8.4.3.6. Columbia Suicide Severity Rating Scale (C-SSRS)

C-SSRS categorization based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories 1, 2, 3, 4, and 7 will be summarized as dichotomous endpoints at End of Study/Early Withdrawal Visits.

### 8.4.4. Interim Analysis

No Interim analyses are planned.

# 8.4.5. Missing Data

There will be no imputation of the missing values. All assessments will be conducted based on all the observed data.

### 9. STUDY CONDUCT

Steps to ensure the accuracy and reliability of data include the selection of qualified investigators and appropriate study sites, review of protocol procedures with the investigator and associated personnel prior to the study, periodic monitoring visits, and meticulous data management.

# 9.1. Sponsor and Investigator Responsibilities

# 9.1.1. Sponsor Responsibilities

The sponsor, and/or sponsor's representative is obligated to conduct the study in accordance with strict ethical principles. The sponsor reserves the right to withdraw a patient from the study, to terminate participation of a study site at any time, and/or to discontinue the study.

The sponsor, or sponsor's representative, agrees to provide the investigator with sufficient material and support to permit the investigator to conduct the study according to the study protocol.

# 9.1.2. Investigator Responsibilities

By signing the Investigator's Agreement, the investigator indicates that she/he has carefully read the protocol, fully understands the requirements, and agrees to conduct the study in accordance with the procedures and requirements described in this protocol.

The investigator also agrees to conduct this study in accordance with all laws, regulations, and guidelines of the pertinent regulatory authorities, including and in accordance with the April 1996 International Conference on Harmonisation (ICH) Guidance for Industry E6 Good Clinical Practice (GCP) and in agreement with the 1996 Version of the Declaration of Helsinki. While delegation of certain aspects of the study to sub-investigators and study coordinators is appropriate, the investigator will remain personally accountable for closely overseeing the study and for ensuring compliance with the protocol and all applicable regulations and guidelines. The investigator is responsible for maintaining a list of all persons that have been delegated study-related responsibilities (e.g., sub-investigators and study coordinators) and their specific study-related duties.

Investigators should ensure that all persons who have been delegated study-related responsibilities are adequately qualified and informed about the protocol, IPs, and their specific duties within the context of the study. Investigators are responsible for providing CRO with documentation of the qualifications, GCP training, and research experience for themselves and their staff as required by the sponsor and the relevant governing authorities.

To ensure compliance with the guidelines, the study will be audited by an independent person. The investigator agrees, by written consent to this protocol, to cooperate fully with compliance checks by allowing access to all study documentation by authorized individuals.

#### 9.2. Site Initiation

Study personnel may not screen or enroll patients into the study until after receiving notification from the sponsor or sponsor's representative that the study can be initiated at the study site. The study site will not be authorized for study initiation until:

- The study site has received the appropriate institutional review board (IRB) approval for the protocol and the appropriate informed consent form (ICF).
- All regulatory documents have been submitted to and approved by the sponsor or sponsor's representative.
- The study site has a clinical trial agreement in place.
- Study site personnel, including the investigator, have participated in a study initiation meeting.

### 9.3. Screen Failures

Patients who fail inclusion and/or exclusion criteria may not be rescreened for the study.

# 9.4. Study Documents

All documentation and material provided by the sponsor, or sponsor's representative for this study are to be retained in a secure location and treated as confidential material.

# 9.4.1. Investigator's Regulatory Documents

The regulatory documents must be received from the investigator and reviewed and approved by the sponsor or sponsor's representative before the study site can initiate the study and before the sponsor, or sponsor's representative, will authorize shipment of investigational product (IP) to the study site. Copies of the investigator's regulatory documents must be retained at the study site in a secure location. Additional documents, including a copy of the protocol and applicable amendment(s), the IB, CRF/electronic case report form (eCRF) completion guidelines, copies of regulatory references, copies of IRB correspondence, and IP accountability records should also be retained as part of the investigator's regulatory documents. It is the investigator's responsibility to ensure that copies of all required regulatory documents are organized, current, and available for inspection.

# 9.4.2. Case Report Forms

By signing the Investigator's Agreement, the investigator agrees to maintain accurate CRFs/eCRFs and source documentation as part of the case histories for all patients who sign an ICF.

Case report forms are considered confidential documents and should be handled and stored accordingly. The sponsor, or sponsor's representative, will provide the necessary training on the use of the specific CRFs/eCRF system used during the study to ensure that the study information is captured accurately and appropriately.

To ensure data accuracy, CRF/eCRF data for individual patient visits should be completed as soon as possible after the visit. All requested information must be entered in the CRF/electronic

data capture (EDC) system according to the completion guidelines provided by the sponsor, or sponsor's representative.

#### 9.4.3. Source Documents

All information recorded in the CRF/EDC system must be supported by corresponding source documentation. Examples of acceptable source documentation include, but are not limited to, hospital records, clinic and office charts, laboratory notes, and recorded data from automated instruments, memoranda, and pharmacy dispensing records.

During the study, select CRF/eCRF data may be used as original data collection tools as long as a description of this documentation process is maintained in the investigator's study files.

Clinical laboratory data required by the protocol will be electronically transferred from the central laboratory to the sponsor or the sponsor's representative. A paper copy of the laboratory results will be provided to the study site and should be retained with each patient's source data.

The investigator will provide direct access to source data and documents for trial-related monitoring, audits, IEC/IRB review, and regulatory requirements.

# 9.5. Study Termination

The study may be terminated at the sponsor's discretion at any time and for any reason. Study sites may be asked to have all patients currently participating in the study complete all of the assessments for the telephone follow-up call.

In the event of study discontinuation, study sites may be asked to have all patients currently participating in the study complete all of the assessments for the Early Withdrawal Visit.

# 9.6. Study Site Closure

At the end of the study, all study sites will be closed. The sponsor or sponsor's representative may terminate participation of a study site at any time. Examples of conditions that may require premature termination of a study site include, but are not limited to, the following:

- Noncompliance with the protocol and/or applicable regulations and guidelines
- Inadequate patient enrollment

### 9.6.1. Record Retention

The investigator shall retain and preserve one copy of all data generated during the course of the study, specifically including, but not limited to, those defined by GCP as essential until the following occur:

- At least 2 years after the last marketing authorization for the Investigational Product has been approved or the sponsor has discontinued its research with the Investigational Product, or
- At least 2 years have elapsed since the formal discontinuation of clinical development of the Investigational Product

These documents should be retained for a longer period, however, if required by the applicable regulatory requirement(s) or if needed by the sponsor.

# 9.6.2. Laboratory Sample Retention

Laboratory samples may be used for purposes related to this research. The samples will be stored until the sponsor has determined that specimens are no longer needed and the decision has been made that none of the samples needs to be reanalyzed. In addition, identifiable samples can be destroyed at any time at the request of the patient.



# 10. QUALITY CONTROL AND QUALITY ASSURANCE

The sponsor or its designee will implement and maintain quality control and quality assurance procedures with written standard operating procedures to ensure the study is conducted and data are generated, documented, and reported in compliance with the protocol, GCP, and applicable regulatory requirements. This trial will be conducted in accordance with the provisions of the Declaration of Helsinki (October 1996) and all revisions thereof, and in accordance with the FDA CFR 312.50 and 312.56, and with the ICH guidelines on GCP (CPMP/ICH/135/95).

### **10.1.** Changes To The Protocol

Only Insys may modify the protocol. Amendments to the protocol will be made only after consultation and agreement between the sponsor and the investigator. The only exception is when the investigator assesses a patient's safety will be compromised without immediate action. In these circumstances, immediate approval of the chairman of the IEC/IRB must be sought, and the investigator should inform the sponsor and the full IEC/IRB within 5 working days after the emergency occurred. All amendments that have an impact on patient risk or the study objectives, or require revision of the informed consent form, must receive approval from the IEC/IRB prior to their implementation.

# 10.2. Monitoring

The sponsor or sponsor's representative will conduct site visits to monitor the study and ensure compliance with the protocol, GCP, and applicable regulations and guidelines. The assigned clinical research associate(s) (CRA[s]) will visit the investigator and study site at periodic intervals and maintain periodic communication. The investigator agrees to allow the CRA(s) and other authorized sponsor/contract research organization (CRO) personnel access. The CRA(s) will maintain current personal knowledge of the study through observation, review of study records and source documentation, and discussion of the conduct of the study with the investigator and staff.

# 10.3. Data Review Meeting

The sponsor will review all data reported in CRFs of all patients before database lock. The data review meeting determines whether all enrolled patients can be included in the analysis population according to the specified definition of analysis populations and evaluates whether or not medical decisions of the investigator were appropriate for important data affecting the safety endpoints.

#### 10.4. Protocol Violations

The investigator will conduct the study in compliance with the protocol approved by the IRB. Modifications to the protocol should not be performed without agreement of both the investigator and the sponsor. Changes to the protocol will require written IRB approval prior to implementation, except when the modification is needed to eliminate an immediate hazard(s) to patients.

The investigator or sub-investigator should document any deviation from the protocol and the reason. If the investigator performs a deviation from the protocol or a change of the protocol to

eliminate an immediate hazard(s) to patients, the record should be immediately submitted to the sponsor, the CRU, and the IRB by the investigator and the IRB will provide expedited review and approval. After the investigator has obtained approval of the IRB, the investigator should obtain written permission of the CRU and written agreement of the sponsor.

When deviation from the protocol is required to eliminate immediate hazard(s) to patients, the investigator will contact the sponsor, if circumstances permit, to discuss the planned course of action. Any deviations from the protocol must be fully documented in the CRF and source documentation.

# 10.5. Quality Assurance Audit

This study will be subject to audit by the sponsor, CRO, or designee.

The sponsor or sponsor's representative may conduct audits on a selection of study sites, requiring access to patient notes, study documentation, and facilities or laboratories used for the study.

The study site, facilities, all data (including source data), and documentation will be made available for audit by quality assurance auditors and for IRB or regulatory authorities according to GCP guidelines. The investigator agrees to cooperate with the auditor during the visit and will be available to supply the auditor with CRFs or other files necessary to conduct that audit. Any findings will be strictly confidential.

If a regulatory authority informs the investigator that it intends to conduct an inspection, the investigator shall notify sponsor or sponsor's representative immediately.

#### 11. REGULATORY AND ETHICAL CONSIDERATIONS

### 11.1. Regulatory Authority Approval

The investigator will ensure that the protocol and consent form are reviewed and approved by the appropriate Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to the start of any study procedures. The IEC/IRB will be appropriately constituted and will perform its functions in accordance with Food and Drug Administration (FDA) regulations, International Conference on Harmonization (ICH) good clinical practice (GCP) guidelines, and local requirements as applicable.

In addition, the IRB will approve all protocol amendments (except for logistical or administrative changes), written informed consent documents and document updates, patient recruitment procedures, written information to be provided to the patients, available safety information, information about payment and compensation available to patients, the investigator's curriculum vitae and/or other evidence of qualifications, and any other documents requested by the IRB/IEC and regulatory authority, as applicable.

# 11.2. Ethical Conduct of the Study

The study will be conducted in accordance with the Declaration of Helsinki and GCP according to ICH guidelines. Specifically, the study will be conducted under a protocol reviewed by an IRB or IEC; the study will be conducted by scientifically and medically qualified persons; the benefits of the study are in proportion to the risks; the rights and welfare of the patients will be respected; the physicians conducting the study do not find the hazards to outweigh the potential benefits; and each patient will give his or her written, informed consent before any protocoldriven tests or evaluations are performed.

# 11.3. Statement of Investigator/Delegation of Authority

As a condition for conducting the clinical investigation, the Principal Investigator will sign the FDA Form 1572, Statement of Investigator (21 Code of Federal Regulations [CFR] Part 312).

The Principal Investigator will ensure that all persons assisting with the trial are adequately qualified, informed about the protocol, any amendments to the protocol, the study treatments, and their trial-related duties and functions. The qualified investigator will maintain a list of sub-investigator and other appropriately qualified persons to whom to delegate significant trial-related duties. Should the qualified investigator delegate the supervision of the investigational product administration to a designated person, this individual must have the appropriate medical qualifications to effectively conduct or supervise any potential resuscitation procedures.

#### 11.4. Patient Informed Consent

The investigator or his/her designee will inform the patient of all aspects pertaining to their participation in the study. The process for obtaining patient informed consent will be in accordance with all applicable regulatory requirements (e.g., CFR Part 50 and ICH E6 Section 4.8). The investigator or his/her designee and the patient must both sign and date the informed consent document (ICD) before they can participate in the study. The patient will receive a copy of the signed and dated form, and the original will be retained in the site's study records. The decision to participate in the study that is made by the patient is entirely voluntary. The

investigator or his/her designee must emphasize to the patient that consent for study participation may be withdrawn at any time without penalty or loss of benefits to which the patient is otherwise entitled. If the ICD is amended during the study the investigator must follow all applicable regulatory requirements pertaining to approval of the amended ICD by the IRB, and use of the amended form, including the necessity of re-consenting ongoing patients.

#### 11.4.1. Assent Guidance

The IRB/IEC must determine, to the extent required by 45 CFR 46.116, that adequate provisions are made for soliciting the assent of pediatric patients (when the IRB/IEC judges that they are capable of providing assent), as well as the permission of the parents (45 CFR 46.408). Permission means the agreement of parent(s) or guardian to the participation of their child or ward in research (45 CFR 46.402(c)). Local and regional/state regulations will also be addressed as applicable.

If the IRB/IEC determines that the capability of some or all of the children is so limited that they cannot reasonably be consulted regarding assent, or that the intervention or procedure involved in the research holds out a prospect of direct benefit that is important to the health or well-being of the children, and is available only in the context of the research, the assent of the children is not a necessary condition for proceeding with the research. Even where the IRB/IEC determines that the patients are capable of assenting, the IRB/IEC may still waive the assent requirement under certain circumstances in accord with 45 CFR 46.116 and 45 CFR 46.408(a). The IRB/IEC and local regulations will determine the age at which assent of patients in this study will not be required. Informed consent from all parent(s)/caregiver(s) will be required.

# 11.5. Investigator Reporting Requirements

In accordance with applicable local regulatory requirements, the investigator may be obligated to provide periodic safety updates on the conduct of the study at his/her site and notification of study closure to the IRB. Such periodic safety updates and notifications are the responsibility of the investigator and not of Insys or its delegate.

### 12. DATA HANDLING AND RECORD KEEPING

The CRO will be responsible for data management and analysis. The procedures will be specified in the Data Management Plan.

# 12.1. Data Management

The CRO will be responsible for activities associated with the data management of this study. The standard procedures for handling and processing records will be followed per GCP and the CRO's SOPs. A comprehensive Data Management Plan will be developed including a data management overview, database contents, annotated CRF and consistency checks. Study site personnel will be responsible for providing resolutions to all data queries. The investigator will be required to document electronic data review to ensure the accuracy of the corrected and/or clarified data.

# 12.2. Case Report Forms and Source Documents

The CRFs will be supplied by the CRO data management services. The complete CRFs will be reviewed, signed, and dated by the qualified investigator and a copy returned to the Sponsor with the final report.

Source documents are defined as original documents, data, and records. This may include hospital records, clinical and office charts, laboratory data/information, patients' diaries or evaluation checklists, pharmacy dispensing and other records, recorded data from automated instruments, microfiches, photographic negatives, microfilm or magnetic media and/or x rays.

### 12.3. Documentation and Retention of Essential Documents

All documents pertaining to the study, including a copy of the approved protocol, copy of the ICD, completed CRFs, source documents, drug accountability and retention records, and other study related documents will be retained in the permanent archives of the study site. These will be available for inspection at any time by the Sponsor or the FDA. Per 21 CFR 312, record retention for this study is required for a period of two years following the date on which this study agent is approved by the FDA for the marketing purposes that were the subject of this investigation; or, if no application is to be filed or if the application is not approved for such indication, until two years following the date on which the entire study is completed, terminated, or discontinued, and the FDA is notified.

The investigator will provide direct access to source data and documents for trial related monitoring, audits, IEC/IRB review, and regulatory requirements.

#### 12.4. Financial Disclosure

These issues will be addressed in a separate agreement between the sponsor and the investigator.

The US FDA Financial Disclosure by Clinical Investigators (21 Code of Federal Regulations [CFR] 54) regulations require sponsors to obtain certain financial information from investigators participating in covered clinical studies; each investigator and sub-investigator is required to provide the required financial information and to promptly update Insys Development Company, Inc., with any relevant changes to their financial information throughout the course of the clinical

study and for up to one year after its completion. This rule applies to all investigators and sub-investigators participating in covered clinical studies to be submitted to the FDA in support of an application for market approval.



# 13. FACILITIES

| Clinical Laboratory: | Medpace |
|-----------------------|----------------------------------|
| | 5375 Medpace Way |
| | Cincinnati, OH 45227 |
| Data Management: | PRA Health Sciences |
| | 4130 Park Lake Avenue, Suite 400 |
| | Raleigh, NC 27612 |
| Statistical Services: | PRA Health Sciences |
| | 4130 Park Lake Avenue, Suite 400 |
| | Raleigh, NC 27612 |
| Pharmacovigilance: | PRA Health Sciences |
| | 4130 Park Lake Avenue, Suite 400 |
| | Raleigh, NC 27612 |

### 14. USE OF INFORMATION AND PUBLICATION POLICY

#### 14.1. Use of Information

All information concerning Cannabidiol Oral Solution and Insys Development Company's operations, such as Insys' patent applications, formulas, manufacturing processes, basic scientific data, or formulation information, supplied by Insys Development Company and not previously published, is considered confidential information.

This confidential information shall remain the sole property of Insys Development Company, shall not be disclosed to others without the written consent of Insys Development Company, and shall not be used except in the performance of this study.

The investigator will maintain a confidential patient identification code list of all patients enrolled in the study (by name and patient number). This list will be maintained at the site, and will not be retrieved by Insys.

# 14.2. Publication Policy

Insys Development Company, Inc. will retain ownership of all data. All proposed publications based on this study will be subject to the sponsor's approval requirements.

# 15. REFERENCES (AVAILABLE UPON REQUEST)

- 1. Investigator's Brochure for Cannabidiol Oral Solution, Edition 8.0, 05 Oct 2017.
- 2. Cunha JM, Carlini EA, Pereira AE, Ramos OL, Pimentel C, Gagliardi R, et al. Chronic administration of cannabidiol to healthy volunteers and epileptic patients. *Pharmacol*. 1980; 21: 175-185.
- 3. Carlini EA, Cunha JM. Hypnotic and antiepileptic effects of cannabidiol. *J Clin Pharmacol.* 1981; 21: 417S-427S.
- 4. Porter BE, Jacobson C. Report of a parent survey of cannabidiol-enriched cannabis use in pediatric treatment-resistant epilepsy. *Epilepsy Behav.* 2013; 29: 574-577.
- 5. Gedde MM, Maa E. Whole cannabis extract of high concentration cannabidiol may calm seizures in highly refractory pediatric epilepsies. *America Epilepsy Society Meeting* 2013; abstract: 3.300.
- 6. Sponsor's internal documentation of analysis.
- 7. Zuardi AW, Shirakawa I, Finkelfarb E, Karniol IG. Action of cannabidiol on the anxiety and other effects produced by delta 9-THC in normal subjects. *Psychopharmacology* 1982; 76: 245-250.
- 8. Bisogno T, Hanus L, De Petrocellis L, et al. Molecular targets for cannabidiol and its synthetic analogues: effect on vanilloid VR1 receptors and on the cellular uptake and enzymatic hydrolysis of anandamide. *Br J Pharmacol*. 2001; 134: 845-852.
- 9. Kathmann M, Flau K, Redmer A, Trankle C, Schlicker E. Cannabidiol is an allosteric modulator at mu- and delta-opioid receptors. *Naunyn Schmiedebergs Arch Pharmacol*. 2006; 372: 354-361.
- 10. Bornheim LM, Grillo MP. Characterization of cytochrome P450 3A inactivation by cannabidiol: possible involvement of cannabidiol-hydroxyquinone as a P450 inactivator. *Chem Res Toxicol.* 1998; 11: 1209 1216.
- 11. Ryan D, Drysdale AJ, Lafourcade C, Pertwee RG, Platt B. Cannabidiol targets mitochondria to regulate intracellular Ca2+ levels. *J Neurosci.* 2009; 29: 2053-2063.
- 12. Russo EB, Burnett A, Hall B, Parker KK. Agonistic properties of cannabidiol at 5-HT1A receptors. *Neurochem Res.* 2005; 30: 1037-1043.
- 13. Carrier EJ, Auchampach JA, Hillard CJ. Inhibition of an equilibrative nucleoside transporter by cannabidiol: a mechanism of cannabinoid immunosuppression. *Proc Natl Acad Sci US.* 2006; 103: 7895-7900.
- 14. Jones NA, Glyn SE, Akiyama S, et al. Cannabidiol exerts anti-convulsant effects in animal models of temporal lobe and partial seizures. *Seizure*. 2012; 21: 344-352.
- 15. Harvey DJ, Samara E, Mechoulam R. Comparative metabolism of cannabidiol in dog, rat and man. *Pharmacol Biochem Behav*. 1991; 40: 523-532.
- 16. Stout SM, Cimino NM. Exogenous cannabinoids as substrates, inhibitors, and inducers of human drug metabolizing enzymes: a systematic review. *Drug Metab Rev.* 2014 Feb; 46: 86-95.

- 17. Bergamaschi MM, Queiroz RH, Zuardi AW, Crippa JA. Safety and side-effects of cannabidiol, a cannabis sativa constituent. *Curr Drug Saf.* 2011b; 6: 237-249.
- 18. Yamaori S, Ebisawa J, Okushima Y, Yamamoto I, Watanabe K. Potent inhibition of human cytochrome P450 3A isoforms by cannabidiol: role of phenolic hydroxyl groups in the resorcinol moiety. *Life Sci.* 2011; 88: 730-736.
- 19. Yamaori S, Kushihara M, Yamamoto I, Watanabe K. Characterization of major phytocannabinoids, cannabidiol and cannabinol, as isoform-selective and potent inhibitors of human CYP1 enzymes. *Biochem Pharmacol*. 2010; 79: 1691-1698.
- 20. Johannessen SI, Landmark CJ. Antiepileptic drug interactions principles and clinical implications. *Curr Neuropharmacol.* 2010; 8: 254-267.
- 21. Yamaori S, Koeda K, Kushihara M, Hada Y, Yamamoto I, Watanabe K. Comparison in the in vitro inhibitory effects of major phytocannabinoids and polycyclic aromatic hydrocarbons contained in marijuana smoke on cytochrome P450 2C9 activity. *Drug Metab Pharmacokinet*. 2012; 27: 294-300.
- 22. Zhu HJ, Wang JS, Markowitz JS, et al. Characterization of P-glycoprotein inhibition by major cannabinoids from marijuana. *J Pharmacol Exp Ther.* 2006; 317: 850-857.
- 23. Holland ML, Panetta JA, Hoskins JM, Bebawy M, Roufogalis BD, Allen JD, et al. The effects of cannabinoids on P-glycoprotein transport and expression in multidrug resistant cells. *Biochem Pharmacol.* 2006; 71: 1146-1154.
- 24. Carlini EA, Cunha JM. Hypnotic and anti-epileptic effects of cannabidiol. *J Clin Pharmacol.* 1981; 21: 417S-427S.
- 25. Mechoulam R, Hanus L. Cannabidiol: an overview of some chemical and pharmacological aspects. Part I: chemical aspects. *Chem Phys Lipids* 2002; 121: 35-43.
- 26. Massi P, Vaccani A, Ceruti S, Colombo A, Abbracchio MP, Parolaro D. Antitumor effects of cannabidiol, a nonpsychoactive cannabinoid, on human glioma cell lines. *J Pharmacol Exp Ther*. 2004; 308: 838-845.
- 27. Consroe P, Wolkin A. Cannabidiol antiepileptic drug comparisons and interactions in experimentally induced seizures in rats. *J Pharmacol Exp Ther.* 1977; 201: 26-32.
- 28. Zuardi AW, Morais SL, Guimarães FS, Mechoulam R. Antipsychotic effect of cannabidiol. *J Clin Psychiatry* 1995; 56: 485-486.
- 29. Gloss D, Vickrey B. Cannabinoids for epilepsy. *Cochrane Database Syst Rev.* 2014; 5;3: CD009270.
- 30. Consroe P, Laguna J, Allender J, et al. Controlled clinical trial of cannabidiol in Huntington's disease. *Pharmacol Biochem Behav.* 1991; 40: 701-708.
- 31. Zuardi AW, Cosme RA, Graeff FG, Guimarães FS. Effects of ipsapirone and cannabidiol on human experimental anxiety. *J Psychopharmacol*. 1993a; 7: 82-88.
- 32. Borgwardt SJ, Allen P, Bhattacharyya S, et al. Neural basis of delta-9-tetrahydrocannabinol and cannabidiol: effects during response inhibition. *Biol Psychiatry*. 2008; 64: 966-973.

- 33. Zuardi AW. Cannabidiol: from an inactive cannabinoid to a drug with wide spectrum of action. *Rev Bras Psiquiatr*. 2008; 30: 271-280.
- 34. Gong H Jr, Tashkin DP, Simmons MS, Calvarese B, Shapiro BJ. Acute and subacute bronchial effects of oral cannabinoids. *Clin Pharmacol and Ther.* 1984; 35: 26-32.
- 35. Zuardi AW, Hallak JE, Dursun SM, et al. Cannabidiol monotherapy for treatment-resistant schizophrenia. *J Psychopharmacol.* 2006; 20: 683-686.
- 36. Zuardi A, Crippa J, Dursun S, Morais S, Vilela J, Sanches R, et al. Cannabidiol was ineffective for manic episode of bipolar affective disorder. *J Psychopharmacol*. 2010; 24: 135-137.
- 37. Glauser TA, Cnaan A, Shinnar S, et al. Ethosuximide, valproic acid, and lamotrigine in childhood absence epilepsy. *N Engl J. Med.* 2010; 362: 790-799.
- 38. Devinsky O, Marsh E, Friedman D, et al. Cannabidiol in subjects with treatment-resistant epilepsy: an open-label interventional trial. *Lancet Neurol*. 2016; 15: 270-8.
- 39. Braut-Boucher F, Braemer R, Bolline A, Kremers P. Comparative toxicological investigation of cannabidiol using two different cell culture systems. *Eur J Cell Biol*. 1986; 42: CT 17 (abstract).
- 40. Devinsky O, Cilio MR, Cross H, Fernandez-Ruiz J, French J, Hill C et al. Cannabidiol: pharmacology and potential therapeutic role in epilepsy and other neuropsychiatric disorders. *Epilepsia* 2014; 55: 791–802.

### 16. INVESTIGATOR SIGNATURE PAGE

| TITLE: | AM | ulticen | ter, | Ope | n-Label, | Flexible | e Dos | se S | Stud | y to | Assess | the |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| IIILLL. | - | - | ~ | · . | C D1 | . • | 1 ~ | 4 | $\sim$ | . 1 | . • | |

Long-Term Safety of Pharmaceutical Grade Synthetic

Cannabidiol Oral Solution in Pediatric Patients with Treatment-

Resistant Childhood Absence Seizures

PROTOCOL NUMBER: INS011-17-113

**PHASE OF STUDY:** Phase 2 Long-Term Safety Study

**PROTOCOL DATE:** 23 Aug 2018

**STUDY SPONSOR:** Insys Development Company, Inc.

1333 South Spectrum Blvd, Suite 100

Chandler, AZ 85286

#### PRINCIPAL INVESTIGATOR COMMITMENT:

I, the undersigned Principal Investigator, submit this statement of commitment as evidence that I understand my responsibilities pursuant to the Code of Federal Regulations (21 CFR § 312.60 through § 312.70, 21 CFR § 11, 50, 54, 56) and ICH E6 Good Clinical Practice guidelines, as well as with any and all applicable federal, state and/or local laws and regulations, and agree to conduct the study in accordance with the protocol referenced herein.

| Principal Investigator Printed Name | - |
|-------------------------------------|------|
| Principal Investigator Signature | Date |